## **Supplement 1: Study Protocol**

Supplement 1 contains the ACTS clinical trial protocol v2.4. In addition, the published clinical trial protocol and statistical analysis plan can be found: *Moskowitz A, Yankama T, Andersen LW for the ACTS Clinical Trial Investigators, et al Ascorbic Acid, Corticosteroids and Thiamine in Sepsis (ACTS) protocol and statistical analysis plan: a prospective, multicentre, double-blind, randomised, placebo-controlled clinical trial BMJ Open 2019;9:e034406.* All analyses were performed as described in the published statistical analysis plan unless otherwise noted in the manuscript.

Supplement 1 additionally contains the original clinical trial protocol in addition to a summary of changes made over time.

| 45 | PROTOCOL V2.4 |
|---|---|
| 46 | |
| 47<br>48 | Ascorbic Acid, Hydrocortisone, and Thiamine in Sepsis and Septic Shock |
| 46<br>49 | A Randomized, Double-Blind, Placebo-Controlled Trial |
| 50 | |
| 51 | Acronym: Ascorbic acid, Corticosteroids, and Thiamine in Sepsis (ACTS) Trial |
| 52 | CLINICAL TRIAL PROTOCOL |
| 53<br>54 | CLINICAL TRIAL PROTOCOL |
| 55 | Version 2.4 |
| 56 | December 13, 2018 |
| 57 | IND: 136882 |
| 58 | |
| 59 | Oliminal Trials Cov. Idoutifican NOT02200555 |
| 60 | Clinical Trials.Gov Identifier: NCT03389555 |
| 61<br>62 | Principal investigator: |
| 63 | Michael W. Donnino, MD |
| 64 | Director of Center for Resuscitation Science |
| 65 | Associate Professor of Medicine, Harvard Medical School |
| 66 | Attending Physician in Emergency and Critical Care Medicine, BIDMC |
| 67 | Dath Land Danier Mathed Oaster |
| 68 | Beth Israel Deaconess Medical Center West Clinical Compus 2 <sup>nd</sup> Floor |
| 69<br>70 | West Clinical Campus 2 <sup>nd</sup> Floor<br>One Deaconess Road, Boston MA 02215 |
| 70<br>71 | Phone: 617-754-2295 |
| 72 | Fax: 617-754-2350 |
| 73 | Email: mdonnino@bidmc.harvard.edu |
| 74 | |
| 75 | Funded By: |
| 76 | Open Philanthropy Project (https://www.openphilanthropy.org/) |
| 77<br>78 | |
| 79 | |
| 80<br>81 | |
| 82 | |
| 83<br>84 | |
| 85 | |
| 86 | |
| 87 | |

| 89<br>90<br>91 | SYNOPSIS | 6 |
|---|---|---|
| 92 | TRIAL OVERVIEW | 7 |
| 93 | STEERING COMMITTEE | 8 |
| 94 | TRIAL SITES | 9 |
| 95 | 1. BACKGROUND AND SIGNIFICANCE | 10 |
| 96 | 1.1 Scope of the Problem | 10 |
| 97 | 1.2 Existing Interventions | 10 |
| 98 | 1.3 The combination of vitamin C, hydrocortisone, and vitamin B1 may improve outcomes | 10 |
| 99 | 1.4 Physiologic Rationale | 10 |
| 100 | 2. TRIAL DESIGN | 11 |
| 101 | 2.1 Overview | 11 |
| 102 | 2.2 Allocation | 11 |
| 103 | 2.3 Intervention | 11 |
| 104 | 2.3.1 Vitamin C, Hydrocortisone, and Vitamin B1 | 11 |
| 105 | 2.3.2 Placebo | 11 |
| 106 | 2.4 Blinding | 11 |
| 107 | 2.5 Regulatory Issues | 11 |
| 108 | 3. SETTING AND PARTICIPANT POPULATION | 12 |
| 109 | 3.1 Setting | 12 |
| 110 | 3.2 Inclusion criteria | 12 |
| 111 | 3.3 Exclusion criteria | 12 |
| 112 | 3.4 Pregnancy | 12 |
| 113 | 4. TRIAL PROCEDURES | 13 |
| 114 | 4.1 Participant Identification | 13 |
| 115 | 4.2 Consent procedures | 13 |
| 116 | 4.3 Randomization | 13 |
| 117 | 4.4 Drug preparation and administration | 13 |
| 118 | 4.4.1 Contingencies and Participant Withdrawal | 14 |
| 119 | 4.5 Specimen collection procedures | 14 |
| 120 | 4.5.1 Timing and volume of blood draw | 14 |
| 121 | 4.5.2 Specimen samples | 14 |
| 122 | 4.5.3 Biomarker tube initial processing and shipping | 15 |
| 123 | 4.6 Study flow diagram | 15 |

| 124 | 4.7 General Sepsis Management | 15 |
|-----|----------------------------------------------------------|----|
| 125 | 4.8 Glucometer use during the study period | 15 |
| 126 | 5. OUTCOMES | 16 |
| 127 | 5.1 Definitions | 16 |
| 128 | 5.1.1 Primary Outcome | 16 |
| 129 | 5.1.2 Key Secondary Outcomes | 16 |
| 130 | 5.2 Rationale for Outcomes | 17 |
| 131 | 5.3 Additional Secondary Outcomes | 17 |
| 132 | 5.3.1 Additional secondary outcomes | 17 |
| 133 | 5.3.2 90-day follow-up for Quality of Life assessment | 17 |
| 134 | 5.4 Safety | 18 |
| 135 | 5.4.1 Definitions | 18 |
| 136 | 5.4.2 Specific adverse event data collection | 18 |
| 137 | 5.4.3 Adverse Event Reporting | 18 |
| 138 | 5.4.5 Safety Monitoring Labs | 19 |
| 139 | 6. SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS PLAN | 19 |
| 140 | 6.1 Sample size calculation | 19 |
| 141 | 6.2 Statistical analysis plan | 20 |
| 142 | 6.2.1 General considerations | 20 |
| 143 | 6.2.2 SOFA score and renal failure | 20 |
| 144 | 6.2.3 30-day mortality | 20 |
| 145 | 6.2.5 Subgroup analyses | 21 |
| 146 | 6.2.6 Statistical stopping criteria | 21 |
| 147 | 7. DATA COLLECTION AND MANAGEMENT | 21 |
| 148 | 7.1 Data collection process | 21 |
| 149 | 7.2 Variables | 21 |
| 150 | 7.3 Data quality and validity | 21 |
| 151 | 7.4 Data storage and security | 21 |
| 152 | 8. ETHICAL CONSIDERATIONS | 22 |
| 153 | 8.1 Risks and Benefits | 22 |
| 154 | 8.1.1 Potential benefits | 22 |
| 155 | 8.1.2 Potential harms | 22 |
| 156 | 9. MONITORING | 23 |
| 157 | 9.1 Institutional Review Board (IRB) | 23 |
| 158 | 9.2 Data Safety and Monitoring Board (DSMB) | 23 |

| 159 | 10 CLINICAL MONITORING PLAN | 24 |
|-----|--------------------------------|----|
| 160 | 11. TIMELINE AND ENROLLMENT | 25 |
| 161 | 11.1 Timeline | 25 |
| 162 | 11.2 Screening & Enrollment | 25 |
| 163 | 12. FUNDING | 26 |
| 164 | 13. PUBLICATION | 26 |
| 165 | 14. DATA SHARING | 26 |
| 166 | 15. TASKS AND RESPONSIBILITIES | |
| 167 | References | |
| 168 | Appendices | |
| 169 | Appendix 1: Abbreviations | |
| 170 | Appendix 2: CAM-ICU Form | 33 |
| 171 | | |

### SYNOPSIS

 The "Ascorbic Acid, Corticosteroids, and Thiamine in Sepsis (ACTS)" trial is a multi-center, double-blind, randomized clinical trial that aims to determine the impact of Vitamin C, Hydrocortisone, and Vitamin B1 vs. Placebo on organ injury and mortality on participants with sepsis and septic shock. The trial will be conducted in accordance with all applicable national and international laws, regulations, and guidelines The trial and this protocol is developed in accordance with the International Conference on Harmonization (ICH) guidelines 1-3 and the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) statement 4.5. The principal investigator wrote the protocol with input from the steering committee. Any substantial changes or amendments to the protocol will be clearly documented and communicated to all relevant parties.

Title

Vitamin C, Hydrocortisone, and Vitamin B1 in Sepsis and Septic Shock – A Randomized, Double-Blind, Placebo-Controlled Trial (The ACTS Trial)

| Clinical Trials Number | NCT03389555 |
|---|---|
| Sources of monetary or material support | Open Philanthropy Project (https://www.openphilanthropy.org/) |
| Study Sites | 12-sites in the United States |
| Condition studied | Sepsis and septic shock |
| Interventions | Vitamin C (1.5g every 6 hours x 4-days), hydrocortisone (50mg every 6 hours x 4-days), and Vitamin B1 (100mg every 6 hours x 4-days) |
| Comparator | Placebo |
| Inclusion criteria | <ul> <li>Adult participant (age ≥ 18 years)</li> <li>Suspected (cultures drawn and antibiotic given) or confirmed (via culture results) infection</li> <li>Receiving vasopressor (norepinephrine, phenylephrine, epinephrine, dopamine, vasopressin, or angiotensin II)</li> </ul> |
| Exclusion criteria | <ul> <li>Member of a protected population (pregnant, prisoner)</li> <li>Known history of kidney stones within the past 1 year</li> <li>End stage renal disease (ESRD) requiring dialysis</li> <li>Known history of G6PD deficiency</li> <li>Known history of Hemochromatosis</li> <li>Comfort Measures Only status</li> <li>Anticipated death within 24-hours despite maximal therapy (as determined by the enrolling physician)</li> <li>Receiving supplemental vitamin B1 in a dose greater than that contained in a multivitamin (&lt;2mg)</li> <li>Clinical indication for steroids (e.g. chronic use) as determined by the clinical team providing this drug</li> <li>Clinical indication for vitamin B1 as determined by the clinical team providing this drug</li> <li>Known allergy to vitamin C, hydrocortisone, or vitamin B1</li> </ul> |
| Study type | Interventional Allocation: Randomized (1:1) Intervention model: Parallel group Masking: Double-blind |
| Target sample size | 200 Participants (100/arm) |
| Primary outcome | Change in the Sequential Organ Failure Assessment (SOFA) score between enrollment and 72-hours |
| Key secondary outcomes | Incidence of renal failure during index ICU stay 30-day mortality |

### STEERING COMMITTEE

### 186 187

### Michael Donnino, M.D.

Associate Professor of Medicine Director, Center for Resuscitation Science Beth Israel Deaconess Medical Center Harvard Medical School

### Ari Moskowitz, M.D.

Attending, Pulmonary and Critical Care Medicine Beth Israel Deaconess Medical Center Harvard Medical School

### Lars W. Andersen, M.D., MPH, Ph.D

Associate Professor of Medicine Research Center for Emergency Medicine Department of Clinical Medicine Aarhus University and Aarhus University Hospital

### Michael N. Cocchi, MD

Assistant Professor of Emergency Medicine Beth Israel Deaconess Medical Center Harvard Medical School

### Paul E. Marik, M.D.\*

Professor of Medicine Chief, Division of Pulmonary and Critical Care Medicine Eastern Virginia Medical School

### Katherine Berg, M.D.

Assistant Professor of Medicine Beth Israel Deaconess Medical Center Harvard Medical School

### Anne Grossestreuer, Ph.D.

Instructor in Emergency Medicine Beth Israel Deaconess Medical Center Harvard Medical School

### Joseph Miller, MD

Attending, Emergency Medicine Department of Emergency Medicine Henry Ford Hospital

### 188 Conflicts of interest

The members of the steering committee have no financial conflicts of interest related to the current trial.

190 191 192

189

\*Stepped down from Steering Committee prior to publication. Was not a site investigator.

### **TRIAL SITES**

<u>Coordinating Center</u> Beth Israel Deaconess Medical Center

330 Brookline Avenue

Boston, MA 02215

Site Investigator: Michael W. Donnino, MD

### **Enrolling Sites\***

| Hospital Name | Location | Site Principal Investigator |
|---|---|---|
| Henry Ford Hospital | Detroit, MI | Junior Uduman, MD |
| DMC-Detroit Receiving Hospital | Detroit, MI | Rob Sherwin, MD |
| DMC-Sinai-Grace Hospital | Detroit, MI | Rob Sherwin, MD |
| Harper Hospital | Detroit, MI | Rob Sherwin, MD |
| UT Health, The University of Texas<br>Health Science Center | Houston, TX | Pratik Doshi, MD |
| Mayo Clinic | Phoenix, AZ | Ayan Sen, MD |
| Beth Israel Deaconess Medical<br>Center | Boston, MA | Ari Moskowitz, MD |
| Beaumont Hospital | Royal Oak, MI | Ron Otero, MD |
| • | , | Kon Otero, MD |
| Brigham and Women's Hospital | Boston, MA | Peter Hou, MD |
| Long Island Jewish Hospital Center - Queens | New York, NY | Maksim Korotun, MD; Jonathan Gong, MD |
| Long Island Jewish Hospital Center – Hyde Park | New York, NY | Ayelet Hilewitz, MD; Jonathan Gong, MD |
| Mount Auburn Hospital | Cambridge, MA | Jessica McCannon, MD |
| University of Pittsburgh | Pittsburgh, PA | David Huang, MD |
| South Shore Hospital | Weymouth, MA | Mark Hershey, MD |

\*Depending on study progress, sites may be added or removed in the future.

### 1. BACKGROUND AND SIGNIFICANCE

### 1.1 Scope of the Problem

The worldwide incidence of sepsis has been estimated at more than 23 million cases<sup>6</sup> and sepsis contributes to more than a third of all hospital deaths in the United States.<sup>7,8</sup> Mortality for those in septic shock with elevated lactate is more than 40%.<sup>9</sup> In addition to high short-term mortality, sepsis is associated with significant post-discharge morbidity and mortality.<sup>10-15</sup> The economic burden for participants suffering from sepsis is staggering with an estimated yearly financial burden of \$17 billion.<sup>16</sup> Treatments are generally limited to antibiotics and intravenous fluids while providing support to maintain organ function.<sup>17,18</sup>

**1.2 E** 

### 1.2 Existing Interventions

To date, numerous interventions have been tested for participants with sepsis and septic shock with limited, if any, success. 19-22 Recently, three large studies found no benefit from early goal directed therapy over usual care in emergency department participants with sepsis. 23-25 Other recent studies focusing on hemodynamics, fluid therapy, and transfusions have also failed to show a significant benefit in this participant population. Previous studies focusing on immunomodulary therapies or drotrecogin alfa have likewise shown disappointing results. 29-35

# **1.3 The combination of vitamin C, hydrocortisone, and vitamin B1 may improve outcomes** In a before-and-after study exploring the effects of the combination of vitamin C, hydrocortisone, and vitamin B1 in a cohort of participants with sepsis and septic shock, Marik et. al. found a remarkable improvement in time to shock reversal ( $18.3 \pm 9.8$ hours vs. $54.9 \pm 28.4$ hours), organ injury ( $\Delta$ SOFA $4.8 \pm 2.4$ vs. $0.9 \pm 2.7$ ), and mortality (8.5% vs. 40.4%) following implementation of the drug 'cocktail' as compared to before implementation even after adjusting for potential confounders. This study joins other promising trials of individual elements of this drug combination. In a trial of vitamin B1 in septic shock, there was a substantial reduction in mortality and organ injury (particularly kidney injury) in those with vitamin B1 deficiency and septic shock who were given vitamin B1 as compared to placebo. In addition, several studies of vitamin C alone have shown promise in critically ill populations and a recent meta-analysis of corticosteroids in sepsis suggests potential benefit.

### 1.4 Physiologic Rationale

The combination of vitamin C, hydrocortisone, and vitamin B1 is hypothesized to improve outcomes in sepsis through a number of mechanisms.<sup>36</sup> Vitamin C is an important contributor to endothelial integrity and severe deficiency states (e.g. scurvy) can result in endothelial breakdown with resultant vascular leak and edema.<sup>44,45</sup> In addition, vitamin C is a potent anti-oxidant and is integral to endogenous vasopressor synthesis.<sup>36</sup> Hydrocortisone, a potential adjunctive therapy in septic shock<sup>46,47</sup>, may act synergistically with vitamin C.<sup>48,49</sup> Vitamin B1, a key cofactor of pyruvate dehydrogenase, is a critical component of metabolic dysfunction without which a shift towards anaerobic energy production occurs.<sup>50</sup> Vitamin B1 is also a necessary component of the pentose phosphate pathway, which plays a role in reducing oxidative stress.<sup>51,52</sup> While the physiologic effects of these drugs given in combination is not entirely known, we hypothesize that there will be synergistic effects with respect the metabolic resuscitation of sepsis.

### 2. TRIAL DESIGN

### 2.1 Overview

This will be an investigator-initiated, multicenter, randomized, placebo-controlled, parallel group, double-blind, superiority trial of vitamin C, hydrocortisone, and vitamin B1 vs. placebo in participants with sepsis and septic shock. A total of 200 adult participants will be enrolled. The primary outcome will be the change in SOFA score between enrollment and 72-hours. Key secondary outcomes include the incidence of renal failure during the index ICU stay and survival at 30 days.

# **2.2 Allocation**

Participants will be randomized in a 1:1 ratio to either the combination of vitamin C, hydrocortisone, and vitamin B1 or placebo in blocks with random sizes of 2 or 4. The randomization will be stratified according to site. <sup>53</sup> An independent statistician will create the randomization list using a random number generator. The complete list will only be shared with an independent pharmacy consultant, who will not be involved in clinical care. The pharmacy consultant and the independent statistician will both store the randomization list. The research pharmacy at each enrolling site will receive a site-specific randomization list.

### 2.3 Intervention

2.3.1 Vitamin C, Hydrocortisone, and Vitamin B1

The study drugs will consist of vitamin C (1.5g every 6 hours x 4-days), hydrocortisone (50mg every 6 hours x 4-days), and vitamin B1 (100mg every 6 hours x 4-days).

### 2.3.2 Placebo

The placebo will consist of matching volumes of normal saline (0.9% NaCl). See below section 4.4 for specifics of drug and placebo preparation.

### 2.4 Blinding

The trial will be double-blind; participants, investigators, and the clinical team will be blinded to the allocation. Only the pharmacy providing the study drug will be aware of the allocation. The pharmacy will not be involved with clinical care or outcome evaluation.

As vitamin C possess a yellow tinge, the bags containing the vitamin C/placebo will be covered with light-protective bags. In testing, after dilution there is not distinguishing characteristics of the vitamin C vs. placebo in the IV tubing. Vitamin C, hydrocortisone, and vitamin B1 are not known to have distinctive rapid effects which could lead to unblinding.

The decision to unblind will be at the complete discretion of the treating physician and clinical team. If a clinical team wishes to unblind a participant (e.g. if anaphylaxis occurs), they will contact the research pharmacy who will reveal the study group to the clinical team (but the research team will remain blinded). However, we do not expect many scenarios where emergency unblinding will be necessary. In case unblinding occurs, the reason(s) will be clearly documented in the case report form. The patient will no longer receive study medications, but will be followed for outcomes.

### 2.5 Regulatory Issues

An Investigational New Drug (IND) application was submitted to and approved by the Food and Drug Administration (FDA) for the study of vitamin C, hydrocortisone, and vitamin B1 in sepsis and septic shock (IND # 136882).

The trial has been registered on ClinicalTrials.gov: NCT03389555

### 3. SETTING AND PARTICIPANT POPULATION

### 3.1 Setting

The trial will be conducted at approximately 13 hospitals in the United States. Additional sites might be recruited if needed.

### 3.2 Inclusion criteria

Inclusion criteria:

- 1) Adult participant (age ≥ 18 years)
- 2) Suspected (cultures drawn and antibiotic given) or confirmed (via culture results) infection
- 3) Receiving (continuous infusion) vasopressor (norepinephrine, phenylephrine, epinephrine, dopamine, angiotensin II, or vasopressin)
  - a. Hypotension related primarily to sepsis as opposed to another cause of hypotension (e.g. bleed, cardiogenic shock)

### 3.3 Exclusion criteria

Exclusion criteria:

- 1) Member of a protected population (pregnant, prisoner)
- 2) Known history of kidney stones within the past 1 year (not including incidentally noted stones noted on imaging studies)
- 3) End stage renal disease requiring dialysis (hemodialysis or peritoneal dialysis)
- 4) Known history of G6PD deficiency
- 5) Known history of Hemochromatosis
- 6) Comfort Measures Only status
- 7) Anticipated death within 24-hours despite maximal therapy (as determined by the enrolling physician)
- 8) Receiving supplemental vitamin B1 in a dose greater than that contained in a multivitamin (<2mg)
- 9) Clinical indication for steroids (e.g. chronic use) as determined by the clinical team providing this drug
- 10) Clinical indication for ascorbic acid supplementation in any form
- 11) Clinical indication for vitamin B1 as determined by the clinical team providing this drug
- 12) Known allergy to vitamin C, hydrocortisone, or vitamin B1

<u>Justification of Inclusion and Exclusion Criteria:</u> The inclusion criteria were chosen to isolate a septic participant population with high risk of organ injury and death. The exclusion criteria were chosen to minimize the risk of potential harm and to ensure that participants enrolled do not already have chronic end-stage renal failure with a high likelihood of early need for renal replacement therapy. By evaluating this high-risk population (i.e., most likely to die), we will target those most likely to benefit and therefore increase the probability of showing efficacy.<sup>19</sup>

### 3.4 Pregnancy

Hydrocortisone is considered pregnancy class C on the basis of animal studies showing an association between prenatal parenteral hydrocortisone use and risk of cleft-palate. In addition, there are concerns about effects of hydrocortisone on fetal growth and the possibility of neonatal adrenal insufficiency. The effects of high-dose vitamin C and thiamine in pregnancy are not entirely known. As such, participants who are pregnant will be excluded from the study. Prior to enrollment, all participants of potentially child-bearing potential (women aged <45 years<sup>54</sup>) will be required to have a negative serum or urine HCG test (generally performed as standard-of-care).

We will additionally inform all women of child-bearing potential who are randomized in this study that we recommend they remain abstinent or use two forms of birth control during the study period and for a period of 48-hours after the last dose of study drug.

### 4. TRIAL PROCEDURES

### 4.1 Participant Identification

Screening will be performed in the emergency department and intensive care units (ICUs) with the assistance of electronic screening mechanisms. Detailed screening logs, with reason(s) for exclusion will be kept at each site and reported in the final publication.

We anticipate that all patients, as part of standard-of-care for the septic patient, will have a urine or serum HCG test performed (if a female of child-bearing age). If this test is not sent as part of standard-of-care, it should be sent prior to consent.

### 4.2 Consent procedures

Informed, written consent will be obtained for all participants prior to enrollment.

 After it is determined that they meet all inclusion criteria and no exclusion criteria, the participant (or legally authorized representative [LAR] if the participant is not able to provide consent) will be approached for written informed consent by a physician co-investigator from the team. The investigator will provide the participant/representative information regarding the background and significance of the study, eligibility criteria, and a description of the protocol. To ensure we are correctly identifying the potential participant's LAR, we communicate with members of the clinical team. The consent process may need to be modified based on site-specific IRB recommendations.

The name of the study investigator obtaining consent will be clearly documented, and this person will sign the informed consent document and provide the date and time of their signature. If a physician is performing remote consent, then a copy of the consent form will be signed as soon as he/she is physically present. Signed copies of the consent form will be given to the participant/surrogate, and the original consent document will be stored in the secure study file. In obtaining and documenting informed consent, each investigator will comply with the applicable regulatory requirements and adhere to the ethical and Good Clinical Practice principles that have their origin in the Declaration of Helsinki.

### 4.3 Randomization

After consent is obtained, the research team will notify the local research pharmacy. The research pharmacy will be in possession of the randomization list and will determine which arm (intervention vs. placebo) the participant will be enrolled in.

Patients should be randomized, consented, and enrolled in the study as soon as possible after meeting inclusion criteria. Patients should not be *consented* if it has been >24hours since the patient met inclusion criteria (i.e. start of vasopressors). At the time of randomization and study drug administration, the patient should still be receiving a vasopressor. The patient should not be given study drug if the vasopressor has been stopped (e.g. patient met inclusion criteria overnight but could not be consented for logistical reasons and then improves to the point of no longer requiring a vasopressor). In this scenario, the paitent will be entered into the dabase as consented but not enrolled.

### 4.4 Drug preparation and administration

The vitamin C and vitamin B1 will be mixed together in 100ml of normal saline and administered intravenously over 45-60 minutes. The hydrocortisone will be given intravenously as a push-dose in 1ml of saline over 1-2 minutes. The placebo will be given using techniques and volumes matching those of the study medications.

All study medications will be continued for 4-days or until the participant expires or leaves the intensive care unit.

### 4.4.1 Contingencies and Participant Withdrawal

- In the unlikely event that a participant is discharged alive from the hospital prior to 4 days after enrollment, all study medications will be stopped. The participant will remain in the study and will be followed for outcomes.
- Hydrocortisone is occasionally used for refractory septic shock. If the clinical team opts to provide a
  participant hydrocortisone, the hydrocortisone will be given open-label but the vitamin C/B1 will
  remain randomized and blinded. In this case, the research team will ensure that study
  hydrocortisone/placebo is replaced by open-label hydrocortisone. The participant will remain in
  the study and will be followed for outcomes.
- If the clinical team decides to give the participant vitamin B1 for clinical purposes, the study drug will be continued (including thiamine) as long as the total maximum dose of vitamin B1 is ≤1,500mg/day. 1,500mg day is a standard dose for Wernicke's encephalopathy at many institutions and has not been associated with any increased harm.
- If the clinical team decides to give the participant vitamin C for clinical purposes, further administration of study meds will be stopped. The participant will remain in the study and will be followed for outcomes.
- If a participant withdraws from the study, further administration of study meds will be stopped. Data collected prior to withdrawal will be maintained but additional data will not be collected.

### 4.5 Specimen collection procedures

4.5.1 Timing and volume of blood draw

All participants will have a blood samples collected at four time-points and urine samples at two time-points (if not already available as part of routine clinical care). Blood will be obtained by venipuncture, or from an existing venous or arterial catheter. Urine will be collected via clean catch urine or via catheter.

### Specimen Collection Time Points

- 1. T1=0 hrs (just before study drug administration)
- 450 2. T2=24 hrs (+/- 2 hrs)
- 451 3. T3=72 hrs (+/- 2 hrs)
- 452 4. T4=120hrs (+/- 12hrs)

### 4.5.2 Specimen samples

At the T1, T2, T3, and T4 time points, blood will be sent for complete blood count (including hemoglobin, white blood cell count, platelet count), a serum chemistry (including sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatining, glucose, aspartate transaminase, alanine transaminase, and total bilirubin), and a venous blood gas to measure lactate. These tests will be performed by the clinical laboratory at each site. As many of these laboratory tests are commonly obtained for clinical purposes, these tests do not need to be repeated if a result is available from the clinical care of the participant within 2 hours of the time point (or within 12 hours of the T4 time-point).

In addition to traditional clinical markers, blood will be obtained for future biomarker analysis (including inflammatory biomarkers, markers of endothelial function, and markers of mitochondrial function), and measurement of vitamin C, vitamin B1, and cortisol levels. The total volume of blood that may be drawn for a participant at each time point will not exceed 60mls. Levels of vitamin C, vitamin B1, and cortisol will be measured at time T1 and time T3 only. 20ml of urine will be collected for future biomarker analysis at T1, T2, and T3.

If performed as part of standard-of-care, results of urinalysis and urine sediment testing will be collected prior to enrollment.

### 4.5.3 Biomarker tube initial processing and shipping

Please see accompanying blood collection standard operating procedure for full details. In brief, 15ml of blood will be drawn into EDTA tubes and 10ml of blood will be drawn into a corvac tube. From one of the EDTA tubes, 3ml of whole blood will be initially drawn and separated into 3x 1ml aliquots. Plasma will then be isolated from the EDTA tube(s) and aliquoted into cryovials as follows: 4x 0.5ml aliquots and the remainder in 1ml aliquots. Serum will then be isolated from the corvac tube, and separated into 1ml aliquots. Cryovials will be protected from light and frozen at -80°C until processing. An additional 20ml of urine will also be collected, centrifuged, and separated into 1ml aliquots then frozen at -80°C until processing.

Sites will be expected to ship frozen samples to the coordinating center after every 5 enrollments. The coordinating center will assist with all shipping procedures.

### 4.6 Study flow diagram



### 4.7 General Sepsis Management

Investigators should follow local sepsis management guidelines. No specific sepsis bundle is required by this study, however the early administration of antibiotics, maintenance of a mean arterial pressure ≥65mmHg with a combination of volume resuscitation and vasopressors, and early source control are recommended—as detailed in the Suriving Sepsis Guidelines.<sup>55</sup> Elements of sepsis care should be reported on the online case report form (CRF).

### 4.8 Glucometer use during the study period

High dose vitamin C has been shown to falsely elevate glucose level readings when measured with certain point-of-care glucometers employing glucosedehydrogenase-pyrroloquinoline quinone amperometric methods<sup>56</sup>. Some commonly used glucometer brands using this approach include Accu-Chek (Roche Diagnostic) and Optium (Abbott Diabetes Care) (but not StatStrip; Nova Biomedical). While the effects of high-dose vitamin C on glucometer readings have been seen primarily at higher doses of vitamin C than are intended for use in this trial,<sup>56</sup> we recommend that sites explore what glocumeters are in use in local ICUs. If locally used glucometers may be

impacted by high serum concentrations of vitamin C (as determined by the manufacturer), we recommend that clinical teams caring for enrolled participants be alerted to the possibility of falsely elevated blood-glucose levels when measured by glucometer. If there is a clinical concern about a glucose reading obtained via glucometer, a serum glucose should be obtained which will not be impacted by vitamin C. In the event of an emergency related to suspected hypoglycemia, glucose should be immediately given while a serum glucose level is pending.

### 5. OUTCOMES

### **5.1 Definitions**

### 5.1.1 Primary Outcome

The primary outcome will be the absolute change in the Sequential Organ Failure Assessment (SOFA]) score from enrollment (time=0) to 72 hours after drug administration. The SOFA score will be defined using a modification in which the SaO2/FiO2 ratio is substituted for the PaO2/FiO2 ratio as has been previously described. <sup>57,58</sup> This modified score will be used so that participants without an existing arterial catheter can be spared arterial puncture.

| Points | SaO2*/FiO2 <sup>§</sup> | Blood Pressure | GCS" | Bilirubin (mg/dL) | Creatinine<br>(mg/dL) | Platelets<br>(x10 <sup>3</sup> µL) |
|---|---|---|---|---|---|---|
| 1 | <400 | < 70 mm/Hg | 13–<br>14 | 1.2–1.9 | 1.2 – 1.9 | <150 |
| 2 | <326 | dopamine ≤ 5 μg/kg/min or<br>dobutamine<br>(any dose) | 10–<br>12 | 2–5.9 | 2.0 – 3.4 | <100 |
| 3 | <236 (and receiving invasive or non-invasive mechanical ventilation) | dopamine > 5µg/kg/min,<br>epinephrine/norepinephrine<br>≤ 0.1 µg/kg/min | 6–9 | 6–11.9 | 3.5 – 4.9<br>Or<br>UOP <sup>†</sup> <500ml/day | <50 |
| 4 | <151(and receiving invasive or non-invasive mechanical ventilation) | dopamine > 15,<br>epinephrine/norepinephrine<br>> 0.1 µg/kg/min | <6 | >12 | > 5.0<br>UOP <sup>†</sup> <200ml/day<br>Or receiving<br>renal<br>replacement<br>therapy | <20 |

\*SaO2=Oxygen saturation (%); § = Fraction of inspired oxygen (%); I = Glasgow Coma Scale; † = Urine Output Fio2 will be determined by using either the set FiO2 (for patients receiving invasive or non-invasive mechanical ventilation) or by adding 3% FiO2 for each liter/minute of supplemental oxygen added up to 100% FiO2 (for patients not receiving mechanical ventilation). Patients with an SaO2/FiO2 ratio <236 who are not receiving invasive or non-invasive mechanical ventilation, will be assigned a score of 2.

### 5.1.2 Key Secondary Outcomes

<u>Incidence of Acute Renal Failure</u> – Renal failure will be defined as the development of Kidney Disease Improving Global Outcomes [KDIGO] Stage 3 acute kidney injury during the index ICU stay after study enrollment.<sup>58</sup>

| KDIGO Stage | Serum creatinine criteria | Urine output criteria |
|---|---|---|
| 1 | Increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.4 µmol/l) or increase to more than or equal to 150% to 200% (1.5-to 2-fold) from baseline | Less than 0.5 ml/kg per hour for more than 6 hours |
| 2 | Increase in serum creatinine to more than 200% to 300% (> 2- to 3- fold) from baseline | Less than 0.5 ml/kg per hour for more than 12 hours |
| 3 | Increase in serum creatinine to more than 300% (> 3-fold) from baseline (or serum creatinine of | Less than 0.3 ml/kg per hour for 24 hours or anuria for 12 hours OR |

| 354 µmol/l] with an acute (RRT) increase of at least 0.5 mg/dl [44 µmol/l]) |
|-----------------------------------------------------------------------------|
|-----------------------------------------------------------------------------|

<u>30-Day Mortality</u> – Mortality at 30-days. This will be assessed by review of the medical records if the participant remains in the hospital or if the participant expired while in the hospital. If the participant was discharged, 30-day mortality will be assessed by contacting the participant by phone or by searching the National Center for Health Statistics (NCHS) National Death Index (NDI) consistent with a recent multicenter phase III trial in sepsis.<sup>23</sup> Phone calls will be made by the research team at each site.

### **5.2 Rationale for Outcomes**

**Change in SOFA score:** Organ failure is highly associated with mortality<sup>60</sup> and improvement in organ function is a key goal for critical care physicians. In the study by Marik et al.<sup>36</sup>, participants who received the 3-drug regimen had substantial improvements in the trajectory of organ failure over the first 72-hours of their ICU stay. If the combination of vitamin C, hydrocortisone, and vitamin B1 can improve organ function in the first 72-hours following ICU admission, we believe that clinicians will likely quickly adopt this safe and inexpensive therapy. Importantly, this outcome can be measured early in the hospital stay and is therefore less likely to be affected by other potential elements of hospital care that can affect more distal outcomes (e.g., mortality).

**Kidney Injury:** Renal failure has been estimated to occur in 23% of participants with sepsis and over 50% of participants with septic shock. In studies of participants with septic shock, there is a step-wise increase in mortality with worsening acute kidney injury (AKI). In addition, many participants who experience renal injury during septic shock do not recover renal function prior to hospital discharge and may require long term dialysis. As both data from the study by Marik et. al. and a separate study of vitamin B1 in septic shock have shown substantial improvements in renal outcomes, kidney failure is a natural secondary outcome and one that could change practice independently from other factors – in other words, many clinicians would likely provide this therapy if they knew that kidney function could be protected, since this organ is vital to long-term health.

**Mortality:** Finally, we will measure 30-day mortality. We anticipate that the combination of vitamin C, hydrocortisone, and vitamin B1 will reduce mortality in this high-risk population.

### **5.3 Additional Secondary Outcomes**

5.3.1 Additional secondary outcomes

Additional secondary outcomes will include length of ICU stay, length of hospital stay, ventilator-free days over the first 7-days after enrollment, shock-free days over the first 7-days after enrollment, and the incidence of delirium on day #3 of the ICU stay (as assessed using the Confusion Assessment Method [CAM-ICU] system). Sites at which the CAM-ICU is performed daily as part of standard-of-care should assess whether delirium occurs on any day during the initial ICU stay. See Appendix #2.

### 5.3.2 90-day follow-up for Quality of Life assessment

Sites may choose to participate in a long-term outcomes substudy exploring the effects of ascorbic acid, hydrocortisone, and thiamine vs. placebo on quality of life following sepsis. If a site chooses to participate, a trained research assistant/investigator at the site (who is blinded to treatment arm) will contact all participants who were alive at 30-days, and perform the SF-36 at day 90 following enrollment. The SF-36 is a 36-Item Short-Form Health Survey (SF-36), a validated survey of general quality of life in adults, can be administered in person or over the telephone by research

personnel. It measures eight different dimensions: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions, as well as one question asking about perceived changes in health. The telephone version of the 36-Item Short-Form Health Survey has been validated and used in sepsis. 66-69

### 5.4 Safety

### 5.4.1 Definitions

The following definitions will be used<sup>70</sup>:

<u>Adverse event</u>: any untoward medical occurrence in a participant to whom a medicinal product is administered and which does not necessarily have a causal relationship with this treatment

<u>Serious adverse event</u>: any untoward medical occurrence that at any dose requires inparticipant hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, results in a congenital anomaly or birth defect, is life-threatening, or results in death

<u>Unexpected serious adverse event</u>: a serious adverse reaction, the nature, severity or outcome of which is not consistent with the reference safety information

### 5.4.2 Specific adverse event data collection

To assess specific amd potentially serious adverse events that may be related to the combination of the study medications, we will collect data on the following:

| Serious Adverse Event | Definition |
|---|---|
| Hyperglycemia | Serum glucose >300mg/dl in the first 120-hours after |
| | enrollment |
| Hypernatremia | Serum sodium (> 150 mmol/L) occurring in the first 120- |
| | hours after enrollment |
| New Infection | A - data-main address the main aireal investigation at a sale |
| Catheter-site | As determined by the site principal investigator at each site. Should be a new organism or site of infection and |
| Lung | believed to be unrelated to the initial presenting |
| Gastrointestinal | infectious source. Many will have the initiation of new |
| Urinary tract | antibiotics or a change in antibiotics. |
| Other | antibiotics of a change in antibiotics. |
| Serious allergic reaction | Anaphylaxis or other allergic reaction requiring systemic |
| | corticosteroids. Allergic reaction should be related (or |
| | suspected to be related) to the study medicaiton |
| Renal calculus | Development of a renal calculus between enrollment |
| | and 30-day follow-up (based on question asked during |
| | follow-up phone call). |

### 5.4.3 Adverse Event Reporting

All unexpected serious adverse events thought to be related to the study drug, and any unexpected fatal or life-threatening adverse events thought to be related to the study drug will be recorded in the online CRF, reported directly to the coordinating center, and reported to the appropriate IRB shortly following the event per local protocol. In addition, unexpected serious adverse events related to the study drug will be undergo expedited reporting to the DSMB within 7 days of the coordinating center becoming aware of the event. The DSMB will additionally review all adverse events in aggregate after every 50 patients are enrolled.

Adverse events will additionally be reported to the FDA as outlined in 21CFR312.32 and summarized below:

- a. All unexpected fatal or life-threatening adverse events thought to be related to the study drug will be reported to the FDA within 7 calendar-days of when the ACTS team is made aware of the event.
- b. All unexpected serious adverse events thought to be related to the study drug will be reported to the FDA within 15 calendar-days of when the ACTS team is made aware.
- c. All serious unexpected adverse events, and any unexpected fatal or life-threatening events thought to be related to the study drug, will be reported back to all site investigators within 15 calendar-days of the event.
- d. The ACTS team will periodically review all published information relating to the safety of each element of the drug combination. Any concerning safety information obtained from this review, or otherwise obtained (e.g. from unpublished scientific papers), will be reported to the FDA within 15 calendar-days.

### 5.4.5 Safety Monitoring Labs

As detailed above, safety monitoring labs will be obtained at 120-hours, after completion of the study protocol.

### 6. SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS PLAN

### 6.1 Sample size calculation

The study has been powered to have at least 80% power for the primary outcome and all key secondary outcomes as follows:

**SOFA Score**: Based on preliminary data<sup>36</sup>, we conservatively anticipate a decrease in SOFA score of 6 (standard deviation [SD]: 4) in the treatment group and 4 (SD: 2) in the placebo group. With these estimates, enrollment of **200 participants (100/arm)** at an alpha of 0.05 and using a t-test with unequal variance, the trial will provide > 99% power to detect a statistical significant difference between groups.

**Kidney Injury:** Based on preliminary data from our study of vitamin B1 in septic shock,<sup>38</sup> we anticipate that 30% of participants in the treatment group and 55% in the placebo group will have renal failure which will result in a 94% power for this outcome. This calculation and following calculation were performed using the Fisher's exact test.

**Mortality:** Based on preliminary data<sup>36,37,71</sup>, we anticipate that the control group will have a mortality of 40%. We estimate a treatment effect of 50% (risk ratio: 0.50) resulting in a mortality of 20% in the treatment group. With these estimates, 182 participants will lead to 80% power. To further increase the trial's power and due to potential loss-to-follow-up, we will aim to enroll 200 participants. These estimates are conservative compared to the Marik et al. study which found a treatment effect corresponding to a risk ratio of 0.21 which persisted in adjusted analysis.<sup>36</sup>

### Sample Size Adjustment

If after 100 patients are enrolled, the overall change in SOFA score is less than anticipated in the above power analysis and/or the renal failure event rate or mortality rate is lower than predicted, the enrollment target of 200 patients may be adjusted accordingly so as to improve power for the primary outcome and all key secondary outcomes at the end of the trial period. Specifically, we will aim to maintain  $\geq$ 90% power to detect a 2-point difference in  $\Delta$ SOFA score (using variance seen for the full cohort) and  $\geq$ 80% power to detect a 50% treatement effect on mortality. Whether to increase the study sample size, and the degree of sample size increase, will be decided on by the blinded Steering Committee who will not have access to data stratified by treatment group. The Steering

Committee will take into account logistical and financial considerations when updating the enrollment target.

### 6.2 Statistical analysis plan

### 6.2.1 General considerations

The statistical analyses and reporting will adhere to the CONSORT guidelines.<sup>72,73</sup> All tests will be two-sided, a p-value < 0.05 will be considered significant, and all confidence intervals will have 95% coverage. All analyses will be conducted on a modified intention-to-treat basis only including participants receiving at least the first dose of the study medications. In a double-blind trial, this approach is unbiased while increasing precision.<sup>74</sup> The two groups will be compared in relation to baseline characteristics using descriptive statistics.

The persons conducting the statistical analysis will be blinded to the randomized allocation. Groups will be designated as "A" and "B" until all pre-specified analyses are performed and shared with all authors and the Data Safety Monitoring Board.

### 6.2.2 SOFA score and renal failure

The change in SOFA score will be calculated and compared between groups using the Wilcoxon Rank Sum test (if the change is not normally distributed) or by a t-test if the change is approximately normally distributed. Fisher's exact tests will be used to compare the incidence of renal failure during the index ICU stay.

 If a participant expires prior to the 72-hour time point, SOFA scores will be imputed based on a predefined plan as follows. If a participant expires before 24-hours has elapsed, a 20% increase from baseline will be imputed. If a participant expires between 24-hours and 48-hours, a 15% increase from the 24-hour time point will be imputed. If a participant dies between 48-hours and 72-hours, a 20% increase from the 24-hour time point will be imputed. Sensitivity analyses will be performed using various other imputation techniques. Specifically, we will perform 1) a sensitivity analysis in which the worst possible SOFA score (score of 24) is imputed for those participants who expire, 2) a sentivity analysis in which the last SOFA score for participants who expire will be carried forward, and 3) a sensitivity analyses were chosen to model 'worst-possible' and 'best-possible' scenarios. For the secondary outcome of renal failure, participants who expire during their ICU stay will be assessed to have developed renal failure if they demonstrated any degree of unresolved KDIGO acute kidney injury prior to death. If there was no evidence of acute kidney injury prior to death or if kidney injury had fully resolved, these participants will be assessed as not having developed renal failure.

### 6.2.3 30-day mortality

Survival until 30 days will be analyzed using survival analysis. Participants lost to follow-up will be censored and the censoring will be assumed non-informative. Results will be presented with Kaplan-Meier curves and the groups compared using the log-rank test. Hazard ratios with 95% confidence intervals will be obtained using Cox's proportional hazards models. The proportional hazards assumption will be verified by visual inspection of the Kaplan-Meier curves and statistically by including a product term (i.e. "interaction") between the treatment group variable and the natural logarithm of time in the model. If the proportional hazards assumption is not met, only the Kaplan-Meier curves and the p-value from the log-rank test will be presented.

Adverse events and other binary outcomes will be presented and analyzed like renal failure.

### 6.2.4 Additional Secondary Analyses

Both ICU and hospital length of stay will be compared using Wilcoxon Rank Sum tests. Ventilator and shock free days over the first 7-days after enrollment will likewise be compared using the

Wilcoxon Rank Sum given that the data will likely be not normally distributed. In these latter two analyses, patients who expire prior to 7-days will be assessed to have 0 ventilator or shock free days if they had died while on a ventilator or vasopressor respectively. The incidence of delirium will be compared using the Fisher's exact test. For the quality-of-life outcome (i.e. 90-day SF-36), the primary analysis will only include patients with available data. As a secondary analysis, multiple imputation will be used to estimate SF-36 scores in all patients not known to be dead at 90 -days.

6.2.5 Subgroup analyses

The analysis will include three pre-defined subgroup analyses for the primary and key secondary outcomes according to 1) participants with initially high SOFA scores ( $\geq$ 9). This cut-off was chosen to represent a population with a  $\geq$ 50% predicted likelihood of mortality<sup>78</sup> 2) baseline vitamin B1 deficiency and 3) baseline adrenal insufficiency. We will not plan to perform a subgroup analysis according to vitamin C deficiency, as prior work has shown that the vast majority of participants with septic shock have vitamin C levels below the reference range. Witamin B1 deficiency will be defined as a plasma vitamin B1 level  $\leq$  7 nmol/L as has been previously described. Adrenal insufficiency will be defined as a cortisol level  $\leq$ 10 $\mu$ g/dL. The trial is not powered to detect subgroup differences and these will be considered exploratory and hypothesis generating.

6.2.6 Statistical stopping criteria

Since the primary outcome is not mortality, there will be no formal stopping criteria for efficacy. There will be no predefined stopping criteria for futility since enrollment of the full cohort might allow for detection of efficacy in subgroups or in other outcomes even if the primary outcome is negative.

### 7. DATA COLLECTION AND MANAGEMENT

### 7.1 Data collection process

Data collection will be the responsibility of the individual site investigators with oversite from the trial coordinating center. Most variables (i.e. demographics, sepsis characteristics and laboratory results) will be obtained prospectively from the electronic medical record. 30-day follow-up regarding safety and mortality end-points will be obtained via telephone call post-discharge (unless the participant remains in the hospital at 30-days). Data will be entered directly into the online database software (see below).

7.2 Variables

Will be provided on the online CRF. A PDF version is available upon request.

7.3 Data quality and validity

Data quality and validity will be optimized by using a detailed data dictionary which will be distributed to all sites. Data quality will be monitored both centrally by the coordinating site and locally by each site principal investigator.

7.4 Data storage and security

The database application we will use is REDCap Cloud (https://www.redcapcloud.com/). REDCap Cloud is a professional database that provides a user-friendly interface. The REDCap Cloud data management system is secure, fully compliant with all regulatory guidelines, and includes a complete audit-trail for data entry validation. Through these mechanisms, as well as relevant training for all involved parties, participant confidentiality will be safeguarded. All members of the research team will be required to complete standardized training in REDCap cloud, which will be documented within the software.

The consent form and other trial documents for each participant will initially be stored in a secure, locked place at the individual sites. Participating sites will be responsible for maintaining their own trial documents and study materials (e.g. signed ICFs, site logs etc). Trial documents generated at the Coordinating Center will be maintained the Coordinating Center. Following completion of the

trial, documents will be maintained for a period of at least 2-years at each site per FDA regulations (or longer depending on local IRB guidelines).

### 8. ETHICAL CONSIDERATIONS

### 8.1 Risks and Benefits

8.1.1 Potential benefits

**Potential Benefits to Individual Participant:** Assuming our hypothesis is correct and our results are comparable to those previously published<sup>36</sup>, individual participants enrolled in our study and randomized to the treatment arm will benefit from a better trajectory of organ failure and improved mortality. As many participants who survive an initial episode of sepsis will have a future admission for sepsis, participants participating in this study but randomized to the placebo arm may see a future benefit from knowledge gained.

**Potential Benefits to Society:** Septic shock remains a highly morbid clinical condition for which there is no specific therapy. Our study, assuming our hypothesis is confirmed, will provide strong support for the widespread adoption of vitamin C, corticosteroids, and vitamin B1 for participants with septic shock. This, in turn, will significantly improve participant outcomes and reduce the global burden of death related to septic shock. Thus, even if participants are randomized to the placebo arm, their involvement with this study has tremendous potential benefits for society as whole. If vitamin C, corticosteroids, and vitamin B1 are found to be neutral or harmful (the latter being highly unlikely), society will benefit as the study will likely prevent the widespread dissemination of an ineffective medication combination.

### 8.1.2 Potential harms

### **Study Drug**

Vitamin C – Ascorbic acid is a water-soluble essential vitamin that is safe even at high doses. Nevertheless, adverse effects related to high-dose ascorbic acid have been described. These adverse effects include diarrhea/abdominal bloating, increased oxalate excretion, iron overload in participants with hemochromatosis, and hemolysis in participants with G6PD deficiency. We exclude participants with known renal failure, known G6PD deficiency, or known hemochromatosis to limit these potential risks. We will additionally exclude participants with known allergy to ascorbic acid. Ascorbic acid has additionally been used in at least 3 clinical trials in critically-ill populations without major associated adverse effect. 40-42

Hydrocortisone – Hydrocortisone is a well-established medication for the treatment of refractory shock in sepsis. Some studies (e.g. CORTICUS) have found an increased incidence of secondary infection in participants with septic shock who receive steroids. This finding has not been replicated in other large trials of corticosteroids for sepsis. Additional hypothetical risks to the administration of hydrocortisone to participants with septic shock (e.g. increased gastro-intestinal bleeding, muscle weakness, and delirium) have not been found in clinical trials of corticosteroids in sepsis. In Interest Principal sepsis in the septic shock (e.g. increased gastro-intestinal bleeding, muscle weakness, and delirium) have not been found in clinical trials of corticosteroids in sepsis. In Interest Principal sepsis in the sepsi

Hydrocortisone will not be tapered in this study as prior studies have shown benefit with corticosteroids in septic shock without a taper. <sup>80</sup> In addition, a recent large trial of corticosteroids in septic shock (ADRENAL, NEJM 2018) randomized patients to 7-days of corticosteroids or placebo and did not include a taper. In that trial there was no reported difference in rates of recurrent shock.

 Vitamin B1 – The only potential serious side effect that has been reported from vitamin B1 administration is an extremely rare anaphylactic reaction (1:250,000 cases) and this might not even be of issue with the current manufactured version of vitamin B1 in the United States. The risk of an anaphylactic reaction was associated with a vitamin complex dispensed in Europe, and whether

vitamin B1 was the actual offending agent remains unknown; however, this 0.0004% theoretical chance of an adverse reaction is incredibly low. In a series of 989 participants in the United States who received intravenous vitamin B1, none had an anaphylactic reaction and the only reported side effects were minor consisting of transient local irritation or in one case pruritus (0.093%). Further safety data comes from the clinical use of intravenous vitamin B1 at our coordinating site. At Beth Israel Deaconess Medical Center (BIDMC, coordinating center) vitamin B1 is provided liberally for participants with nutritional deficiency – for example, BIDMC has administered intravenous vitamin B1 in over 8,000 separate participant encounters from 2002 until present. Despite this heavy usage, no adverse reactions were reported in any of the 8,000 participant encounters.

The combination of vitamin C, hydrocortisone and vitamin B1 – To date, the only study of the combination of vitamin C, hydrocortisone and vitamin B1 was the above referenced study by Marik et. al.

 All procedures will take place at the study site. All research procedures and monitoring will be conducted by experienced personnel, and participants will be in the ICU given critical illness. This permits closer observation and more detailed monitoring by clinicians familiar with the care of participants experiencing and resuscitated from septic shock.

### **Blood Collection**

Most participants will have existing venous or arterial catheters in place and we will be able to collect blood from these ports, essentially eliminating the risks associated with blood collection. In the very rare case that a participant does not have an indwelling line, the risk of venipuncture is extremely low, and will not exceed the risk of clinical blood draws the participant will already be receiving.

### **Loss of Confidentiality**

All measures will be taken to ensure that no confidential information is released. All participant information will be stored in a password protected database to which only study investigators will have access. Additionally, all hard copies of study data will be kept in a locked office accessible only to study investigators. Thus, the risk of loss of confidentiality is very low.

### 9. MONITORING

### 9.1 Institutional Review Board (IRB)

The study will be reviewed and approved by the IRB at each participating site.

### 9.2 Data Safety and Monitoring Board (DSMB)

The DSMB will be responsible for safeguarding the interests of trial participants, assessing the safety and efficacy of the interventions during the trial, and for monitoring the overall conduct of the clinical trial. The DSMB will consist of three clinicians with critical care experience in the management of septic participants. An independent biostatistician/epidemiologist will prepare all DSMB reports. The DSMB members will be chosen such to avoid any financial or intellectual conflicts of interest. The DSMB will review deidentified data after every 50 participants are enrolled to assess for safety; unless there are group differences necessitating unblinding (as determined by the DSMB), the DSMB will be blinded to treatment groups. The trial will continue while the DSMB review data. After each review, the DSMB will create a short report to the steering committee with recommendations for continuation, modifications, or termination of the trial. Criteria for recommending termination will be at the discretion of the DSMB and there will be no formal statistical criteria for termination due to efficacy or safety. A detailed charter for the DSMB will be provided.

### **DSMB Members**

Clifton Callaway, MD, PhD 876 University of Pittsburgh 877 400A Iroquois 878 Pittsburgh, PA 15260 879 (412) 647-8287 880 callawaycw@upmc.edu 881 882 Professor (tenured) of Emergency Medicine; Executive Vice-Chair of Emergency Medicine; UPMC Professor of Emergency Medicine Research 883 884 Expertise: Cardiac Arrest/Clinical Trials 885 Taylor Thompson, MD 886 Massachusetts General Hospital 887 55 Fruit Street 888 Boston, MA 02114 889 (617) 724-7823 890 tthompson1@partners.org 891 Professor of Medicine, Harvard Medical School 892 Director, Critical Care Translational Research, Pulmonary/Critical Care Unit, MGH 893 894 Medical Director, ARDS Network Clinical Coordinating Center Expertise: Sepsis/Clinical Trials 895 896 897 Shahzad Shaefi, MD MPH [DSMB Chair] 898 Beth Israel Deaconess Medical Center One Deaconess Raod 899 Boston, MA 02115 900 901 (617) 355-6286 sshaefi@bidmc.harvard.edu 902 Attending Physician, Department of Anesthesia, Critical Care and Pain 903 904 Expertise: Critical Care Medicine 905

The detailed clinical monitoring plan has been developed and is available from the Coordinating

906

907

908

**10 CLINICAL MONITORING PLAN** 

Center upon request.

### 11. TIMELINE AND ENROLLMENT

### 11.1 Timeline



### 11.2 Screening & Enrollment

Enrollment at each site will be continuously monitored by the site investigator and the principal investigator. Each site will be expected to maintain a screening log including all participants who meet all eligibility criteria at that site. A standardized screening log will be provided to each site via RedCap Cloud—thus allowing for continuous updating of the screening log and will allow capture of all screening failures.

Enrollment will be competitive (i.e. without specific enrollment caps). Number of enrollments at each site will be shared with all sites on a monthly basis. Sites will be expected to complete all elements of the online CRF within 48-hours of each time point. In the case that a site continuously underperforms despite troubleshooting and feedback, the steering committee will evaluate whether enrollment will continue at that site.

**12** 

### 12. FUNDING

Funding for the present trial is provided by the Good Ventures Foundation (http://www.goodventures.org/). The funding agency will have no role in the design and conduct of the study, collection, management, analysis, and interpretation of the data, preparation, review, or approval of the manuscript, or the decision to submit the manuscript for publication.

### **13. PUBLICATION**

The manuscript will adhere to the CONSORT guidelines.<sup>72,73</sup> The principal investigator will be responsible for assigning authorship position and will follow authorship guidelines from the International Committee of Medical Journal Editors.<sup>82</sup> At a minimum, all members of the Steering Committee and all site Principal Investigators (for sites enrolling at least 10 participants) will be included in the primary author list. The main results will be presented at an international conference. The trial results will be shared with participating sites and via press releases but not directly with the participants.

### 14. DATA SHARING

Six months after the publication of the last results, all de-identified individual participant data will be made available for data sharing. Brocedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data. There will be no predetermined end date for the data sharing. Data will be available for any research purpose to all interested parties who have approval from an independent ethics review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Interested parties will be able to request the data by contacting the principal investigator. Authorship of publications emerging from the shared data will follow standard authorship guidelines from the International Committee of Medical Journal Editors and might or might not include authors from the steering committee depending on the nature of their involvement.

### 15. TASKS AND RESPONSIBILITIES

<u>Principal investigator and sponsor</u>: Overall responsibility for protocol development, funding, budget overview, data dictionary development, ethical approval, trial registration, daily management, trial oversight and collection of adverse events, contact to the pharmacy, contact to Good Clinical Practice monitoring unit and the data and safety monitoring board, assessment of overall recruitments, potential recruitment of additional sites, data analysis, and dissemination and presentation of results.

<u>Steering committee</u>: Protocol development, funding, budget overview, data dictionary development, trial oversight, dissemination of results, responsibilities as principal investigator for short time periods.

<u>Site investigators</u>: Responsible for site-specific enrollment, evaluation of eligible patients not included, education of personnel at participating sites, reporting of site-specific issues or challenges to the principal investigator, participant consent for data collection, collecting and reporting data regarding adverse drug events.

<u>Clinical team</u>: Administration of the study drug, participant consent for data collection.

### 971 References

- 972 1. ICH Harmonised Tripartite Guideline. Integrated Addendum To ICH E6(R1): Guideline For Good Clinical Practice E6(R2). 2016;
- http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E6/E6\_R2\_\_Step \_\_4.pdf. Accessed June 30, 2017.
- 976 2. ICH Harmonised Tripartite Guideline. General Considerations for Clinical Trials E8. 1997;
- 977 http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E8/Step4/E8\_Guideline.pdf. Accessed June 30, 2017.
- 979 3. ICH Harnomised Tripartite Guidelines. Statistical Principles for Clinical Trials. 1998;
- 980 http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E9/Step4/E9\_Gui deline.pdf. Accessed June 30, 2017.
- 982 4. Chan AW, Tetzlaff JM, Altman DG, et al. SPIRIT 2013 statement: defining standard protocol items for clinical trials. *Ann Intern Med.* 2013;158(3):200-207.
- 5. Chan AW, Tetzlaff JM, Gotzsche PC, et al. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. *BMJ*. 2013;346:e7586.
- 986 6. Fleischmann C, Scherag A, Adhikari N, et al. Global burden of sepsis: a systematic review (abstract).
  987 *Critical Care*. 2015;19 (suppl 1).
- 7. Liu V, Escobar GJ, Greene JD, et al. Hospital deaths in patients with sepsis from 2 independent cohorts. *Jama*. 2014;312(1):90-92.
- 990 8. Cohen J, Vincent JL, Adhikari NK, et al. Sepsis: a roadmap for future research. *The Lancet Infectious diseases*. 2015;15(5):581-614.
- 992 9. Dellinger RP, Levy MM, Rhodes A, et al. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. *Critical care medicine*. 2013;41(2):580-637.
- Yende S, Linde-Zwirble W, Mayr F, Weissfeld LA, Reis S, Angus DC. Risk of cardiovascular events in survivors of severe sepsis. *American journal of respiratory and critical care medicine*.
   2014;189(9):1065-1074.
- 997 11. Mayr FB, Yende S, Angus DC. Epidemiology of severe sepsis. Virulence. 2014;5(1):4-11.
- 998 12. Wintermann GB, Brunkhorst FM, Petrowski K, et al. Stress Disorders Following Prolonged Critical Illness in Survivors of Severe Sepsis. *Critical care medicine*. 2015.
- 1000 13. Goodwin AJ, Rice DA, Simpson KN, Ford DW. Frequency, cost, and risk factors of readmissions among severe sepsis survivors. *Critical care medicine*. 2015;43(4):738-746.
- 1002 14. Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. *Jama*. 2010;304(16):1787-1794.
- 1004 15. Ortego A, Gaieski DF, Fuchs BD, et al. Hospital-based acute care use in survivors of septic shock. 1005 *Critical care medicine.* 2015;43(4):729-737.
- 1006 16. Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. *The New England journal of medicine*. 2003;348(16):1546-1554.
- 1008 17. Gaieski DF, Edwards JM, Kallan MJ, Carr BG. Benchmarking the incidence and mortality of severe sepsis in the United States. *Critical care medicine*. 2013;41(5):1167-1174.
- 1010 18. Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe 1011 sepsis in the United States: analysis of incidence, outcome, and associated costs of care. *Critical care* 1012 *medicine*. 2001;29(7):1303-1310.
- 1013 19. Deans KJ, Haley M, Natanson C, Eichacker PQ, Minneci PC. Novel therapies for sepsis: a review. *The Journal of trauma*. 2005;58(4):867-874.
- Eichacker PQ, Parent C, Kalil A, et al. Risk and the efficacy of antiinflammatory agents: retrospective and confirmatory studies of sepsis. *American journal of respiratory and critical care medicine*.
   2002;166(9):1197-1205.
- 1018 21. Opal SM, Dellinger RP, Vincent JL, Masur H, Angus DC. The next generation of sepsis clinical trial designs: what is next after the demise of recombinant human activated protein C?\*. *Critical care medicine*. 2014;42(7):1714-1721.

- 1021 22. Angus DC. The search for effective therapy for sepsis: back to the drawing board? *Jama*. 2011;306(23):2614-2615.
- ProCess Investigators, Yealy DM, Kellum JA, et al. A randomized trial of protocol-based care for early septic shock. *The New England journal of medicine*. 2014;370(18):1683-1693.
- 1025 24. Investigators A, Group ACT, Peake SL, et al. Goal-directed resuscitation for patients with early septic shock. *The New England journal of medicine*. 2014;371(16):1496-1506.
- 1027 25. Mouncey PR, Osborn TM, Power GS, et al. Trial of early, goal-directed resuscitation for septic shock.
  1028 The New England journal of medicine. 2015;372(14):1301-1311.
- Asfar P, Meziani F, Hamel JF, et al. High versus low blood-pressure target in patients with septic shock. *The New England journal of medicine*. 2014;370(17):1583-1593.
- 1031 27. Caironi P, Tognoni G, Masson S, et al. Albumin replacement in patients with severe sepsis or septic shock. *The New England journal of medicine*. 2014;370(15):1412-1421.
- Holst LB, Haase N, Wetterslev J, et al. Lower versus higher hemoglobin threshold for transfusion in septic shock. *The New England journal of medicine*. 2014;371(15):1381-1391.
- Abraham E, Anzueto A, Gutierrez G, et al. Double-blind randomised controlled trial of monoclonal antibody to human tumour necrosis factor in treatment of septic shock. NORASEPT II Study Group. *Lancet.* 1998;351(9107):929-933.
- 1038 30. Abraham E, Naum C, Bandi V, et al. Efficacy and safety of LY315920Na/S-5920, a selective inhibitor of 14-kDa group IIA secretory phospholipase A2, in patients with suspected sepsis and organ failure.

  1040 Critical care medicine. 2003;31(3):718-728.
- Abraham E, Wunderink R, Silverman H, et al. Efficacy and safety of monoclonal antibody to human tumor necrosis factor alpha in patients with sepsis syndrome. A randomized, controlled, double-blind, multicenter clinical trial. TNF-alpha MAb Sepsis Study Group. *JAMA : the journal of the American Medical Association*. 1995;273(12):934-941.
- Fisher CJ, Jr., Agosti JM, Opal SM, et al. Treatment of septic shock with the tumor necrosis factor receptor:Fc fusion protein. The Soluble TNF Receptor Sepsis Study Group. *The New England journal of medicine*. 1996;334(26):1697-1702.
- Bernard GR, Wheeler AP, Russell JA, et al. The effects of ibuprofen on the physiology and survival of patients with sepsis. The Ibuprofen in Sepsis Study Group. *The New England journal of medicine*. 1997;336(13):912-918.
- Marti-Carvajal AJ, Sola I, Gluud C, Lathyris D, Cardona AF. Human recombinant protein C for severe
   sepsis and septic shock in adult and paediatric patients. *The Cochrane database of systematic* reviews. 2012;12:CD004388.
- 1054 35. Ranieri VM, Thompson BT, Barie PS, et al. Drotrecogin alfa (activated) in adults with septic shock.

  1055 The New England journal of medicine. 2012;366(22):2055-2064.
- Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine
   for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. *Chest*.
   2017;151(6):1229-1238.
- Donnino MW, Andersen LW, Chase M, et al. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. *Crit Care Med.* 2016;44(2):360-367.
- Moskowitz A, Andersen LW, Cocchi MN, Karlsson M, Patel PV, Donnino MW. Thiamine as a Renal Protective Agent in Septic Shock. A Secondary Analysis of a Randomized, Double-Blind, Placebo-controlled Trial. *Annals of the American Thoracic Society*. 2017;14(5):737-741.
- Teng J, Pourmand A, Mazer-Amirshahi M. Vitamin C: The next step in sepsis management? *J Crit Care.* 2017;43:230-234.
- Fowler AA, 3rd, Syed AA, Knowlson S, et al. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. *Journal of translational medicine*. 2014;12:32.

- Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation
   fluid volumes in severely burned patients using ascorbic acid administration: a randomized,
   prospective study. *Archives of surgery (Chicago, III : 1960)*. 2000;135(3):326-331.
- Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's
   requirement in septic shock. *Journal of research in pharmacy practice*. 2016;5(2):94-100.
- 43. Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y. Corticosteroids for treating sepsis.
   1075 Cochrane Database Syst Rev. 2015(12):CD002243.
- 1076 44. May JM, Harrison FE. Role of vitamin C in the function of the vascular endothelium. *Antioxidants & redox signaling.* 2013;19(17):2068-2083.
- Han M, Pendem S, Teh SL, Sukumaran DK, Wu F, Wilson JX. Ascorbate protects endothelial barrier
   function during septic insult: Role of protein phosphatase type 2A. Free radical biology & medicine.
   2010;48(1):128-135.
- Sprung CL, Annane D, Keh D, et al. Hydrocortisone therapy for patients with septic shock. *The New England journal of medicine*. 2008;358(2):111-124.
- Keh D, Trips E, Marx G, et al. Effect of Hydrocortisone on Development of Shock Among Patients
   With Severe Sepsis: The HYPRESS Randomized Clinical Trial. *Jama*. 2016;316(17):1775-1785.
- Okamoto K, Tanaka H, Makino Y, Makino I. Restoration of the glucocorticoid receptor function by the phosphodiester compound of vitamins C and E, EPC-K1 (L-ascorbic acid 2-[3,4-dihydro-2,5,7,8-tetramethyl-2-(4,8,12-trimethyltridecyl)-2H-1-benzopyran-6 -yl hydrogen phosphate] potassium salt), via a redox-dependent mechanism. *Biochemical pharmacology.* 1998;56(1):79-86.
- 49. Fujita I, Hirano J, Itoh N, Nakanishi T, Tanaka K. Dexamethasone induces sodium-dependant vitamin
   1090 C transporter in a mouse osteoblastic cell line MC3T3-E1. *The British journal of nutrition*.
   1091 2001;86(2):145-149.
- Donnino MW, Andersen LW, Chase M, et al. Randomized, Double-Blind, Placebo-Controlled Trial of
   Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. *Critical care medicine*.
   2016;44(2):360-367.
- 1095 51. Gioda CR, de Oliveira Barreto T, Primola-Gomes TN, et al. Cardiac oxidative stress is involved in heart failure induced by thiamine deprivation in rats. *American journal of physiology Heart and circulatory physiology*. 2010;298(6):H2039-2045.
- Pacal L, Tomandl J, Svojanovsky J, et al. Role of thiamine status and genetic variability in transketolase and other pentose phosphate cycle enzymes in the progression of diabetic
   nephropathy. Nephrology, dialysis, transplantation: official publication of the European Dialysis and
   Transplant Association European Renal Association. 2011;26(4):1229-1236.
- 1102 53. Kernan WN, Viscoli CM, Makuch RW, Brass LM, Horwitz RI. Stratified randomization for clinical trials. 1103 *J Clin Epidemiol.* 1999;52(1):19-26.
- Johnson K, Posner SF, Biermann J, et al. Recommendations to improve preconception health and health care--United States. A report of the CDC/ATSDR Preconception Care Work Group and the Select Panel on Preconception Care. MMWR Recommendations and reports: Morbidity and mortality weekly report Recommendations and reports. 2006;55(Rr-6):1-23.
- 1108 55. Rhodes A, Evans LE, Alhazzani W, et al. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. *Critical care medicine*. 2017;45(3):486-552.
- Flannery AH, Bastin MLT, Magee CA, Bensadoun ES. Vitamin C in Sepsis: When It Seems Too Sweet, It Might (Literally) Be. *Chest.* 2017;152(2):450-451.
- 1112 57. Pandharipande PP, Shintani AK, Hagerman HE, et al. Derivation and validation of Spo2/Fio2 ratio to impute for Pao2/Fio2 ratio in the respiratory component of the Sequential Organ Failure Assessment score. *Critical care medicine*. 2009;37(4):1317-1321.
- 1115 58. Grissom CK, Brown SM, Kuttler KG, et al. A modified sequential organ failure assessment score for critical care triage. *Disaster medicine and public health preparedness.* 2010;4(4):277-284.
- 1117 59. Mehta RL, Kellum JA, Shah SV, et al. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. *Critical care (London, England)*. 2007;11(2):R31.

- de Grooth HJ, Geenen IL, Girbes AR, Vincent JL, Parienti JJ, Oudemans-van Straaten HM. SOFA and mortality endpoints in randomized controlled trials: a systematic review and meta-regression analysis. *Crit Care*. 2017;21(1):38.
- 1122 61. Schrier RW, Wang W. Acute renal failure and sepsis. *The New England journal of medicine*. 2004;351(2):159-169.
- 1124 62. Kellum JA, Chawla LS, Keener C, et al. The Effects of Alternative Resuscitation Strategies on Acute
  1125 Kidney Injury in Patients with Septic Shock. *American journal of respiratory and critical care*1126 medicine. 2016;193(3):281-287.
- Ely EW, Inouye SK, Bernard GR, et al. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). *Jama*. 2001;286(21):2703-2710.
- 1130 64. Watson EK, Firman DW, Baade PD, Ring I. Telephone administration of the SF-36 health survey:
  1131 validation studies and population norms for adults in Queensland. *Aust N Z J Public Health*.
  1132 1996;20(4):359-363.
- Garcia M, Rohlfs I, Vila J, et al. Comparison between telephone and self-administration of Short Form Health Survey Questionnaire (SF-36). *Gac Sanit*. 2005;19(6):433-439.
- Schmidt K, Worrack S, Von Korff M, et al. Effect of a Primary Care Management Intervention on
   Mental Health-Related Quality of Life Among Survivors of Sepsis: A Randomized Clinical Trial. *Jama*.
   2016;315(24):2703-2711.
- Dinglas VD, Hopkins RO, Wozniak AW, et al. One-year outcomes of rosuvastatin versus placebo in sepsis-associated acute respiratory distress syndrome: prospective follow-up of SAILS randomised trial. *Thorax.* 2016;71(5):401-410.
- Zhang K, Mao X, Fang Q, et al. Impaired long-term quality of life in survivors of severe sepsis:
   Chinese multicenter study over 6 years. *Anaesthesist*. 2013;62(12):995-1002.
- 1143 69. Wittbrodt P, Haase N, Butowska D, et al. Quality of life and pruritus in patients with severe sepsis
   1144 resuscitated with hydroxyethyl starch long-term follow-up of a randomised trial. *Crit Care*.
   1145 2013;17(2):R58.
- The European Parliament and the Council of the European Unit. Clinical Trials Regulation (CTR) EU No 536/2014. 2014; https://ec.europa.eu/health/sites/health/files/files/eudralex/vol-1/reg\_2014\_536/reg\_2014\_536\_en.pdf. Accessed July 18, 2017.
- 71. Rhee C, Dantes R, Epstein L, et al. Incidence and Trends of Sepsis in US Hospitals Using Clinical vs Claims Data, 2009-2014. *JAMA*. 2017;318(13):1241-1249.
- 1151 72. Schulz KF, Altman DG, Moher D, Group C. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. *BMJ*. 2010;340:c332.
- 1153 73. Moher D, Hopewell S, Schulz KF, et al. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. *BMJ.* 2010;340:c869.
- Fergusson D, Aaron SD, Guyatt G, Hebert P. Post-randomisation exclusions: the intention to treat principle and excluding patients from analysis. *BMJ*. 2002;325(7365):652-654.
- 75. Fleming T, Harrington D. Nonparametric estimation of the survival distribution in censored data.

  \*\*Communications in Statistics Theory and Methods. 1984;13(20):2469–2486.
- 76. Cox D. Regression models and life tables. *Journal of the Royal Statistical Society.* 1972; Series
   B(20):187–220.
- 1161 77. Kleinbaum D, Klein M. Survival Analysis: A Self-Learning Text. 3rd ed: Springer; 2013.
- Vincent JL, de Mendonca A, Cantraine F, et al. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working
- group on "sepsis-related problems" of the European Society of Intensive Care Medicine. *Critical care medicine*. 1998;26(11):1793-1800.
- 1166 79. Levine M, Rumsey SC, Daruwala R, Park JB, Wang Y. Criteria and recommendations for vitamin C intake. *Jama*. 1999;281(15):1415-1423.

| 1168 | 80. | Annane D, Sebille V, Charpentier C, et al. Effect of treatment with low doses of hydrocortisone and |
|---|---|---|
| 1169 | | fludrocortisone on mortality in patients with septic shock. Jama. 2002;288(7):862-871. |

- Wrenn KD, Murphy F, Slovis CM. A toxicity study of parenteral thiamine hydrochloride. *Annals of emergency medicine*. 1989;18(8):867-870.
- 1172 82. International Committee of Medical Journal Editors. Defining the Role of Authors and Contributors.
  1173 2017; http://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role1174 of-authors-and-contributors.html. Accessed July 6, 2017.
- Taichman DB, Sahni P, Pinborg A, et al. Data Sharing Statements for Clinical Trials A Requirement of the International Committee of Medical Journal Editors. *N Engl J Med.* 2017;376(23):2277-2279.

| 1177 | Appendices | |
|---|---|---|
| 1178 | Annondiv 1. A | hhraviationa |
| 1179<br>1180 | Appendix 1: A | International Conference on Harmonization |
| 1180 | | Standard Protocol Items: Recommendations for Interventional Trials |
| 1182 | | Ascorbic Acid, Corticosteroids, and Thiamine |
| 1183 | | End Stage Renal Disease |
| 1184 | | Sequential Organ Failure Assessment |
| 1185 | | Investigational New Drug |
| 1186 | | Food and Drug Administration |
| 1187 | | Intensive Care Unit |
| 1188 | | Oxygen Saturation |
| 1189 | | Fraction of Inspired Oxygen |
| 1190 | | Glasgow Coma Scale |
| 1191 | | Urine Output |
| 1192 | | Renal Replacement Therapy |
| 1193 | | Confusion Assessment Method |
| 1194 | | National Center for Health Statistics |
| 1195 | | National Death Index |
| 1196 | | Acute Kidney Injury |
| 1197 | | tandard deviation |
| 1198 | | Case Report Form |
| 1199 | | Beth Israel Deaconess Medical Center (Coordinating Center) |
| 1200 | | Institutional Review Board |
| 1201 | DSMB | Data Safety and Monitoring Board |
| 1202 | | |
| 1203 | | |
| 1204 | | |
| 1205 | | |
| 1206 | | |
| 1207 | | |
| 1208 | | |
| 1209 | | |
| 1210 | | |
| 1211 | | |
| 1212 | | |
| 1213 | | |
| 1214 | | |
| 1215 | | |
| 1216 | | |
| 1217 | | |
| 1218 | | |
| 1219 | | |
| 1220 | | |
| 1221 | | |
| 1222 | | |
| 1223 | | |
| 1224 | | |

### **CAM-ICU Worksheet**

| Feature 1: Acute Onset or Fluctuating Course | Score | Check here if Present |
|---|---|---|
| Is the pt different than his/her baseline mental status? OR Has the patient had any fluctuation in mental status in the past 24 hours as evidenced by fluctuation on a sedation scale (i.e., RASS), GCS, or previous delirium assessment? | Either question Yes | |
| Feature 2: Inattention | | |
| Letters Attention Test (See training manual for alternate Pictures) | | |
| <u>Directions</u> : Say to the patient, "I am going to read you a series of 10 letters. Whenever you hear the letter 'A,' indicate by squeezing my hand." Read letters from the following letter list in a normal tone 3 seconds apart. | Number of Errors >2 → | |
| SAVEAHAART | | |
| Errors are counted when patient fails to squeeze on the letter "A" and when the patient squeezes on any letter other than "A." | | |
| Feature 3: Altered Level of Consciousness | | |
| Present if the Actual RASS score is anything other than alert and calm (zero) | RASS<br>anything other<br>than zero → | |
| Feature 4:Disorganized Thinking | | |
| Yes/No Questions (See training manual for alternate set of questions) | | |
| 1. Will a stone float on water? 2. Are there fish in the sea? 3. Does one pound weigh more than two pounds? 4. Can you use a hammer to pound a nail? | Combined | |
| Errors are counted when the patient incorrectly answers a question. | number of | |
| Command Say to patient: "Hold up this many fingers" (Hold 2 fingers in front of patient) "Now do the same thing with the other hand" (Do not repeat number of fingers) *If pt is unable to move both arms, for 2 <sup>nd</sup> part of command ask patient to "Add one more finger" | errors >1→ | |
| An error is counted if patient is unable to complete the entire command. | | |

| Overall CAM-ICU | Criteria Met → | CAM-ICU Positive (Delirium Present) |
|---|---|---|
| Feature 1 plus 2 and either 3 or 4 present = CAM-ICU positive | Criteria Not Met → | CAM-ICU |
| | | Negative<br>(No Delirium) |

| 1229 | 2. PROTOCOL V2.1 (ORIGINAL) |
|---|---|
| 1230<br>1231 | Ascorbic Ccid, Hydrocortisone, and Thiamine in Sepsis and Septic Shock – A Randomized, Double-Blind, Placebo-Controlled Trial |
| 1232 | , transcomeda, ecapio emia, riacoso comionos rina. |
| 1233 | Acronym: Ascorbic acid, Corticosteroids, and Thiamine in Sepsis (ACTS) Trial |
| 1234 | Therefore the dela, Controcatore and Trial mile in Copele (TCTC) Than |
| 1235 | CLINICAL TRIAL PROTOCOL |
| 1236 | CEIMICAE TRIAETROTOGOE |
| 1237 | Version 2.1 |
| 1238 | February 2 <sup>nd</sup> , 2018 |
| | IND: 136882 |
| 1239 | IND. 130002 |
| 1240 | |
| 1241 | Olivia de Triala O a del all'Esta NOTOCOCCEE |
| 1242 | Clinical Trials.Gov Identifier: NCT03389555 |
| 1243 | |
| 1244 | Principal investigator: |
| 1245 | Michael W. Donnino, MD |
| 1246 | Director of Center for Resuscitation Science |
| 1247 | Associate Professor of Medicine, Harvard Medical School |
| 1248 | Attending Physician in Emergency and Critical Care Medicine, BIDMC |
| 1249 | |
| 1250 | Beth Israel Deaconess Medical Center |
| 1251 | West Clinical Campus 2 <sup>nd</sup> Floor |
| 1252 | One Deaconess Road, Boston MA 02215 |
| 1253 | Phone: 617-754-2295 |
| 1254 | Fax: 617-754-2350 |
| 1255 | Email: mdonnino@bidmc.harvard.edu |
| 1256 | |
| 1257 | Funded By: |
| 1258 | Open Philanthropy Project (https://www.openphilanthropy.org/) |
| 1259 | |
| 1260 | |
| 1261 | |
| 1262 | |
| 1263 | |
| 1264 | |
| 1265 | |
| 1266 | |
| 1267 | |
| 1268 | |
| 1269 | |
| 1270<br>1271 | |

| 1272 | | |
|---|---|---|
| 1273 | SYNOPSIS | 38 |
| 1274 | TRIAL OVERVIEW | 39 |
| 1275 | STEERING COMMITTEE | 40 |
| 1276 | TRIAL SITES | 41 |
| 1277 | 1. BACKGROUND AND SIGNIFICANCE | 42 |
| 1278 | 1.1 Scope of the Problem | 42 |
| 1279 | 1.2 Existing Interventions | 42 |
| 1280 | 1.3 The combination of vitamin C, hydrocortisone, and vitamin B1 may improve outcomes | 42 |
| 1281 | 1.4 Physiologic Rationale | 42 |
| 1282 | 2. TRIAL DESIGN | 43 |
| 1283 | 2.1 Overview | 43 |
| 1284 | 2.2 Allocation | 43 |
| 1285 | 2.3 Intervention | 43 |
| 1286 | 2.3.1 Vitamin C, Hydrocortisone, and Vitamin B1 | 43 |
| 1287 | 2.3.2 Placebo | 43 |
| 1288 | 2.4 Blinding | 43 |
| 1289 | 2.5 Regulatory Issues | 43 |
| 1290 | 3. SETTING AND PARTICIPANT POPULATION | 44 |
| 1291 | 3.1 Setting | 44 |
| 1292 | 3.2 Inclusion criteria | 44 |
| 1293 | 3.3 Exclusion criteria | 44 |
| 1294 | 3.4 Pregnancy | 44 |
| 1295 | 4. TRIAL PROCEDURES | 45 |
| 1296 | 4.1 Participant Identification | 45 |
| 1297 | 4.2 Consent proecdures | 45 |
| 1298 | 4.3 Randomization | 45 |
| 1299 | 4.4 Drug preparation and administration | 45 |
| 1300 | 4.4.1 Contingencies and Participant Withdrawal | 45 |
| 1301 | 4.5 Specimen collection procedures | 46 |
| 1302 | 4.5.1 Timing and volume of blood draw | 46 |
| 1303 | 4.5.2 Specimen samples | 46 |
| 1304 | 4.5.3 Biomarker tube initial processing and shipping | |
| 1305 | 4.6 Study flow diagram | 47 |
| 1306 | 4.7 General Sepsis Management | 47 |

| 1307 | 4.8 Glucometer use during the study period | 47 |
|------|----------------------------------------------------------|----|
| 1308 | 5. OUTCOMES | 47 |
| 1309 | 5.1 Definitions | 47 |
| 1310 | 5.1.1 Primary Outcome | 47 |
| 1311 | 5.1.2 Key Secondary Outcomes | 48 |
| 1312 | 5.2 Rationale for Outcomes | 48 |
| 1313 | 5.3 Additional Secondary Outcomes | 49 |
| 1314 | 5.3.1 Additional secondary outcomes | 49 |
| 1315 | 5.3.2 90-day follow-up for Quality of Life assessment | 49 |
| 1316 | 5.4 Safety | 49 |
| 1317 | 5.4.1 Definitions | 49 |
| 1318 | 5.4.2 Specific adverse event data collection | 50 |
| 1319 | 5.4.3 Adverse Event Reporting | 50 |
| 1320 | 5.4.5 Safety Monitoring Labs | 50 |
| 1321 | 6. SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS PLAN | 50 |
| 1322 | 6.1 Sample size calculation | 50 |
| 1323 | 6.2 Statistical analysis plan | 51 |
| 1324 | 6.2.1 General considerations | 51 |
| 1325 | 6.2.2 SOFA score and renal failure | 51 |
| 1326 | 6.2.3 30-day mortality | 51 |
| 1327 | 6.2.5 Subgroup analyses | 52 |
| 1328 | 6.2.6 Statistical stopping criteria | 52 |
| 1329 | 7. DATA COLLECTION AND MANAGEMENT | 52 |
| 1330 | 7.1 Data collection process | 52 |
| 1331 | 7.2 Variables | 52 |
| 1332 | 7.3 Data quality and validity | 52 |
| 1333 | 7.4 Data storage and security | 52 |
| 1334 | 8. ETHICAL CONSIDERATIONS | 53 |
| 1335 | 8.1 Risks and Benefits | 53 |
| 1336 | 8.1.1 Potential benefits | 53 |
| 1337 | 8.1.2 Potential harms | 53 |
| 1338 | 9. MONITORING | 54 |
| 1339 | 9.1 Institutional Review Board (IRB) | 54 |
| 1340 | 9.2 Data Safety and Monitoring Board (DSMB) | 54 |
| 1341 | 10 CLINICAL MONITORING PLAN | 55 |
| 1342 | 11. TIMELINE AND ENROLLMENT | 56 |
|------|--------------------------------|----|
| 1343 | 11.1 Timeline | 56 |
| 1344 | 11.2 Screening & Enrollment | 56 |
| 1345 | 12. FUNDING | 57 |
| 1346 | 13. PUBLICATION | 57 |
| 1347 | 14. DATA SHARING | 57 |
| 1348 | 15. TASKS AND RESPONSIBILITIES | 57 |
| 1349 | References | |
| 1350 | Appendices | 63 |
| 1351 | Appendix 1: Abbreviations | 63 |
| 1352 | Appendix 2: CAM-ICU Form | 64 |
| 1353 | | |

### **SYNOPSIS**

 The "Ascorbic Acid, Corticosteroids, and Thiamine in Sepsis (ACTS)" trial is a multi-center, double-blind, randomized clinical trial that aims to determine the impact of Vitamin C, Hydrocortisone, and Vitamin B1 vs. Placebo on organ injury and mortality on participants with sepsis and septic shock. The trial will be conducted in accordance with all applicable national and international laws, regulations, and guidelines The trial and this protocol is developed in accordance with the International Conference on Harmonization (ICH) guidelines 1-3 and the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) statement 4.5. The principal investigator wrote the protocol with input from the steering committee. Any substantial changes or amendments to the protocol will be clearly documented and communicated to all relevant parties.

Title

Vitamin C, Hydrocortisone, and Vitamin B1 in Sepsis and Septic Shock – A Randomized, Double-Blind, Placebo-Controlled Trial (The ACTS Trial)

| Clinical Trials Number | NCT03389555 |
|---|---|
| Sources of monetary or | Open Philanthropy Project |
| material support | (https://www.openphilanthropy.org/) |
| Study Sites | 12-sites in the United States |
| Condition studied | Sepsis and septic shock |
| Interventions | Vitamin C (1.5g every 6 hours x 4-days), hydrocortisone (50mg every 6 hours x 4-days), and Vitamin B1 (100mg every 6 hours x 4-days) |
| Comparator | Placebo |
| Inclusion criteria | Adult participant (age ≥ 18 years) |
| | <ul> <li>Suspected (cultures drawn and antibiotic given) or<br/>confirmed (via culture results) infection</li> <li>Receiving vasopressor (norepinephrine,<br/>phenylephrine, epinephrine, dopamine, vasopressin, or<br/>angiotensin II)</li> </ul> |
| Exclusion criteria | <ul> <li>Member of a protected population (pregnant, prisoner)</li> <li>Known history of kidney stones within the past 1 year</li> <li>Known history of chronic kidney disease (CKD stage ≥3b [GFR &lt; 45ml/hr])</li> <li>Known history of G6PD deficiency</li> <li>Known history of Hemochromatosis</li> <li>Comfort Measures Only status</li> <li>Anticipated death within 24-hours despite maximal therapy (as determined by the enrolling physician)</li> <li>Receiving supplemental vitamin B1 in a dose greater than that contained in a multivitamin (&lt;2mg)</li> <li>Clinical indication for steroids (e.g. chronic use) as determined by the clinical team providing this drug</li> <li>Clinical indication for vitamin B1 as determined by the clinical team providing this drug</li> <li>Known allergy to vitamin C, hydrocortisone, or vitamin B1</li> </ul> |
| Study type | Interventional Allocation: Randomized (1:1) Intervention model: Parallel group Masking: Double-blind |
| Target sample size | 200 Participants (100/arm) |
| Primary outcome | Change in the Sequential Organ Failure Assessment (SOFA) score between enrollment and 72-hours |
| Key secondary outcomes | Incidence of renal failure during index ICU stay 30-day mortality |

#### STEERING COMMITTEE

### 1368 1369

### Michael Donnino, M.D.

Associate Professor of Medicine Director, Center for Resuscitation Science Beth Israel Deaconess Medical Center Harvard Medical School

### Ari Moskowitz, M.D.

Attending, Pulmonary and Critical Care Medicine Beth Israel Deaconess Medical Center Harvard Medical School

### Lars W. Andersen, M.D., MPH, Ph.D

Associate Professor of Medicine Research Center for Emergency Medicine Department of Clinical Medicine Aarhus University and Aarhus University Hospital

### Michael N. Cocchi, MD

Assistant Professor of Emergency Medicine Beth Israel Deaconess Medical Center Harvard Medical School

#### Paul E. Marik, M.D.

Professor of Medicine Chief, Division of Pulmonary and Critical Care Medicine Eastern Virginia Medical School

# Katherine Berg, M.D.

Assistant Professor of Medicine Beth Israel Deaconess Medical Center Harvard Medical School

### Anne Grossestreuer, Ph.D.

Instructor in Emergency Medicine Beth Israel Deaconess Medical Center Harvard Medical School

### Joseph Miller, MD

Attending, Emergency Medicine Department of Emergency Medicine Henry Ford Hospital

#### 1370 Conflicts of interest

The members of the steering committee have no financial conflicts of interest related to the current trial.

#### **TRIAL SITES**

### 

<u>Coordinating Center</u> Beth Israel Deaconess Medical Center

330 Brookline Avenue 

Boston, MA 02215

Site Investigator: Michael W. Donnino, MD

### **Enrolling Sites\***

| Hospital Name | Location | Site Principal Investigator |
|---|---|---|
| Henry Ford Hospital | Detroit, MI | Joseph Miller, MD |
| DMC-Detroit Receiving Hospital | Detroit, MI | Rob Sherwin, MD |
| DMC-Sinai-Grace Hospital | Detroit, MI | Rob Sherwin, MD |
| UT Health, The University of Texas<br>Health Science Center | Houston, TX | Pratik Doshi, MD |
| Mayo Clinic | Phoenix, AZ | Ayan Sen, MD |
| Beth Israel Deaconess Medical<br>Center | Boston, MA | Ari Moskowitz, MD |
| Beaumont Hospital | Royal Oak, MI | Ron Otero, MD |
| Brigham and Women's Hospital | Boston, MA | Peter Hou, MD |
| Long Island Jewish Hospital Center - Queens | New York, NY | Maksim Korotun, MD |
| Long Island Jewish Hospital Center – Hyde Park | New York, NY | Ayelet Hilewitz, MD |
| Mount Auburn Hospital | Cambridge, MA | Jessica McCannon, MD |
| Univerity of Pittsburgh | Pittsburgh, PA | David Huang, MD |

<sup>\*</sup>Depending on study progress, sites may be added or removed in the future.

#### 3. BACKGROUND AND SIGNIFICANCE

### 1.1 Scope of the Problem

 The worldwide incidence of sepsis has been estimated at more than 23 million cases<sup>6</sup> and sepsis contributes to more than a third of all hospital deaths in the United States.<sup>7,8</sup> Mortality for those in septic shock with elevated lactate is more than 40%.<sup>9</sup> In addition to high short-term mortality, sepsis is associated with significant post-discharge morbidity and mortality.<sup>10-15</sup> The economic burden for participants suffering from sepsis is staggering with an estimated yearly financial burden of \$17 billion.<sup>16</sup> Treatments are generally limited to antibiotics and intravenous fluids while providing support to maintain organ function.<sup>17,18</sup>

# 1.2 Existing Interventions

To date, numerous interventions have been tested for participants with sepsis and septic shock with limited, if any, success. 19-22 Recently, three large studies found no benefit from early goal directed therapy over usual care in emergency department participants with sepsis. 23-25 Other recent studies focusing on hemodynamics, fluid therapy, and transfusions have also failed to show a significant benefit in this participant population. 26-28 Previous studies focusing on immunomodulary therapies or drotrecogin alfa have likewise shown disappointing results. 29-35

**1.3 The combination of vitamin C, hydrocortisone, and vitamin B1 may improve outcomes** In a before-and-after study exploring the effects of the combination of vitamin C, hydrocortisone, and vitamin B1 in a cohort of participants with sepsis and septic shock, Marik et. al. found a remarkable improvement in time to shock reversal ( $18.3 \pm 9.8$  hours vs.  $54.9 \pm 28.4$  hours), organ injury ( $\Delta$ SOFA  $4.8 \pm 2.4$  vs.  $0.9 \pm 2.7$ ), and mortality (8.5% vs. 40.4%) following implementation of the drug 'cocktail' as compared to before implementation even after adjusting for potential confounders. This study joins other promising trials of individual elements of this drug combination. In a trial of vitamin B1 in septic shock, there was a substantial reduction in mortality and organ injury (particularly kidney injury) in those with vitamin B1 deficiency and septic shock who were given vitamin B1 as compared to placebo. In addition, several studies of vitamin C alone have shown promise in critically ill populations 39-42 and a recent meta-analysis of corticosteroids in sepsis suggests potential benefit.

### 1.4 Physiologic Rationale

The combination of vitamin C, hydrocortisone, and vitamin B1 is hypothesized to improve outcomes in sepsis through a number of mechanisms.<sup>36</sup> Vitamin C is an important contributor to endothelial integrity and severe deficiency states (e.g. scurvy) can result in endothelial breakdown with resultant vascular leak and edema.<sup>44,45</sup> In addition, vitamin C is a potent anti-oxidant and is integral to endogenous vasopressor synthesis.<sup>36</sup> Hydrocortisone, a potential adjunctive therapy in septic shock<sup>46,47</sup>, may act synergistically with vitamin C.<sup>48,49</sup> Vitamin B1, a key cofactor of pyruvate dehydrogenase, is a critical component of metabolic dysfunction without which a shift towards anaerobic energy production occurs.<sup>50</sup> Vitamin B1 is also a necessary component of the pentose phosphate pathway, which plays a role in reducing oxidative stress.<sup>51,52</sup> While the physiologic effects of these drugs given in combination is not entirely known, we hypothesize that there will be synergistic effects with respect the metabolic resuscitation of sepsis.

#### 1448 4. TRIAL DESIGN

#### 2.1 Overview 1449

- This will be an investigator-initiated, multicenter, randomized, placebo-controlled, parallel group, 1450
- 1451 double-blind, superiority trial of vitamin C, hydrocortisone, and vitamin B1 vs. placebo in participants with sepsis and septic shock. A total of 200 adult participants will be enrolled. The primary outcome 1452
- will be the change in SOFA score between enrollment and 72-hours. Key secondary outcomes 1453
- 1454 include the incidence of renal failure during the index ICU stay and survival at 30 days.

#### 1455 1456 2.2 Allocation

1457

1458

1459

1460 1461

1462 1463

1464

1465

1469

1471

1472 1473 1474

1475

1476

1477 1478 1479

1480

1481

1482 1483 1484

1485

1486

1487

1488

1489 1490 1491

1492

1493

1494 1495 1496

1497 1498 Participants will be randomized in a 1:1 ratio to either the combination of vitamin C, hydrocortisone, and vitamin B1 or placebo in blocks with random sizes of 2 or 4. The randomization will be stratified according to site.<sup>53</sup> An independent statistician will create the randomization list using a random number generator. The complete list will only be shared with an independent pharmacy consultant, who will not be involved in clinical care. The pharmacy consultant and the independent statistician will both store the randomization list. The research pharmacy at each enrolling site will receive a site-specific randomization list.

#### 2.3 Intervention

- 1466 2.3.1 Vitamin C, Hydrocortisone, and Vitamin B1
- The study drugs will consist of vitamin C (1.5g every 6 hours x 4-days), hydrocortisone (50mg every 6 1467 1468 hours x 4-days), and vitamin B1 (100mg every 6 hours x 4-days).

#### 1470 2.3.2 Placebo

The placebo will consist of matching volumes of normal saline (0.9% NaCl). See below section 4.4 for specifics of drug and placebo preparation.

### 2.4 Blinding

The trial will be double-blind; participants, investigators, and the clinical team will be blinded to the allocation. Only the pharmacy providing the study drug will be aware of the allocation. The pharmacy will not be involved with clinical care or outcome evaluation.

As vitamin C possess a yellow tinge, the bags containing the vitamin C/placebo will be covered with light-protective bags. In testing, after dilution there is not distinguishing characteristics of the vitamin C vs. placebo in the IV tubing. Vitamin C, hydrocortisone, and vitamin B1 are not known to have distinctive rapid effects which could lead to unblinding.

The decision to unblind will be at the complete discretion of the treating physician and clinical team. If a clinical team wishes to unblind a participant (e.g. if anaphylaxis occurs), they will contact the research pharmacy who will reveal the study group to the clinical team (but the research team will remain blinded). However, we do not expect many scenarios where emergency unblinding will be necessary. In case unblinding occurs, the reason(s) will be clearly documented in the case report form. The patient will no longer receive study medications, but will be followed for outcomes.

### 4.5 Regulatory Issues

An Investigational New Drug (IND) application was submitted to and approved by the Food and Drug Administration (FDA) for the study of vitamin C, hydrocortisone, and vitamin B1 in sepsis and septic shock (IND # 136882).

The trial has been registered on ClinicalTrials.gov: NCT03389555

#### 1499 3. SETTING AND PARTICIPANT POPULATION

### **3.1 Setting**

The trial will be conducted at 12 hospitals in the United States. Additional sites might be recruited if needed.

#### 3.2 Inclusion criteria

Inclusion criteria:

- 4) Adult participant (age ≥ 18 years)
- 5) Suspected (cultures drawn and antibiotic given) or confirmed (via culture results) infection
- 6) Receiving (continuous infusion) vasopressor (norepinephrine, phenylephrine, epinephrine, dopamine, or vasopressin)

### 3.3 Exclusion criteria

Exclusion criteria:

- 13) Member of a protected population (pregnant, prisoner)
- 14) Known history of kidney stones within the past 1 year (not including incidentally noted stones noted on imaging studies)
- 15) Known history of chronic kidney disease (CKD stage ≥3b [GFR < 45ml/hr])
- 16) Known history of G6PD deficiency
- 17) Known history of Hemochromatosis
- 18) Comfort Measures Only status
- 19) Anticipated death within 24-hours despite maximal therapy (as determined by the enrolling physician)
- 20) Receiving supplemental vitamin B1 in a dose greater than that contained in a multivitamin (<2mg)
- 21) Clinical indication for steroids (e.g. chronic use) as determined by the clinical team providing this drug
- 22) Clinical indication for vitamin B1 as determined by the clinical team providing this drug
- 23) Known allergy to vitamin C, hydrocortisone, or vitamin B1

<u>Justification of Inclusion and Exclusion Criteria:</u> The inclusion criteria were chosen to isolate a septic participant population with high risk of organ injury and death. The exclusion criteria were chosen to minimize the risk of potential harm and to ensure that participants enrolled do not already have chronic end-stage renal failure with a high likelihood of early need for renal replacement therapy. By evaluating this high-risk population (i.e., most likely to die), we will target those most likely to benefit and therefore increase the probability of showing efficacy.<sup>19</sup>

#### 3.4 Pregnancy

Hydrocortisone is considered pregnancy class C on the basis of animal studies showing an association between prenatal parenteral hydrocortisone use and risk of cleft-palate. In addition, there are concerns about effects of hydrocortisone on fetal growth and the possibility of neonatal adrenal insufficiency. The effects of high-dose vitamin C and thiamine in pregnancy are not entirely known. As such, participants who are pregnant will be excluded from the study. Prior to enrollment, all participants of potentially child-bearing potential (women aged <45 years<sup>54</sup>) will be required to have a negative serum or urine HCG test (generally performed as standard-of-care).

We will additionally inform all women of child-bearing potential who are randomized in this study that we recommend they remain abstinent or use two forms of birth control during the study period and for a period of 48-hours after the last dose of study drug.

#### 4. TRIAL PROCEDURES

#### 4.1 Participant Identification

Screening will be performed in the emergency department and intensive care units (ICUs) with the assistance of electronic screening mechanisms. Detailed screening logs, with reason(s) for exclusion will be kept at each site and reported in the final publication.

We anticipate that all patients, as part of standard-of-care for the septic patient, will have a urine or serum HCG test performed (if a female of child-bearing age). If this test is not sent as part of standard-of-care, it should be sent prior to consent.

#### 4.2 Consent proecdures

Informed, written consent will be obtained for all participants prior to enrollment.

After it is determined that they meet all inclusion criteria and no exclusion criteria, the participant (or legally authorized representative [LAR] if the participant is not able to provide consent) will be approached for written informed consent by a physician co-investigator from the team. The investigator will provide the participant/representative information regarding the background and significance of the study, eligibility criteria, and a description of the protocol. To ensure we are correctly identifying the potential participant's LAR, we communicate with members of the clinical team. The consent process may need to be modified based on site-specific IRB recommendations.

The name of the study investigator obtaining consent will be clearly documented, and this person will sign the informed consent document and provide the date and time of their signature. If a physician is performing remote consent, then a copy of the consent form will be signed as soon as he/she is physically present. Signed copies of the consent form will be given to the participant/surrogate, and the original consent document will be stored in the secure study file. In obtaining and documenting informed consent, each investigator will comply with the applicable regulatory requirements and adhere to the ethical and Good Clinical Practice principles that have their origin in the Declaration of Helsinki.

#### 4.3 Randomization

After consent is obtained, the research team will notify the local research pharmacy. The research pharmacy will be in possession of the randomization list and will determine which arm (intervention vs. placebo) the participant will be enrolled in.

### 4.4 Drug preparation and administration

The vitamin C and vitamin B1 will be mixed together in 100ml of normal saline and administered intravenously over 45-60 minutes. The hydrocortisone will be given intravenously as a push-dose in 1ml of saline over 1-2 minutes. The placebo will be given using techniques and volumes matching those of the study medications.

All study medications will be continued for 4-days or until the participant expires or leaves the intensive care unit.

### 4.4.1 Contingencies and Participant Withdrawal

- In the unlikely event that a participant is discharged alive from the hospital prior to 4 days after enrollment, all study medications will be stopped. The participant will remain in the study and will be followed for outcomes.
- Hydrocortisone is occasionally used for refractory septic shock. If the clinical team opts to provide a
  participant hydrocortisone, the hydrocortisone will be given open-label but the vitamin C/B1 will
  remain randomized and blinded. In this case, the research team will ensure that study

- hydrocortisone/placebo is replaced by open-label hydrocortisone. The participant will remain in the study and will be followed for outcomes.
- If the clinical team decides to give the participant either vitamin B1 or vitamin C for clinical purposes, further administration of study meds will be stopped. The participant will remain in the study and will be followed for outcomes.
  - If a participant withdraws from the study, further administration of study meds will be stopped. Data collected prior to withdrawal will be maintained but additional data will not be collected.

### 4.5 Specimen collection procedures

1609 4.5.1 Timing and volume of blood draw

All participants will have a blood samples collected at four time-points and urine samples at two time-points (if not already available as part of routine clinical care). Blood will be obtained by venipuncture, or from an existing venous or arterial catheter. Urine will be collected via clean catch urine or via catheter.

- 1615 Specimen Collection Time Points
- 1616 1. T1=0 hrs (just before study drug administration)
- 1617 2. T2=24 hrs (+/- 2 hrs)
- 1618 3. T3=72 hrs (+/- 2 hrs)
- 1619 4. T4=120hrs (+/- 12hrs)

### 4.5.2 Specimen samples

At the T1, T2, T3, and T4 time points, blood will be sent for complete blood count (including hemoglobin, white blood cell count, platelet count), a serum chemistry (including sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatining, glucose, aspartate transaminase, alanine transaminase, and total bilirubin), and a venous blood gas to measure lactate. These tests will be performed by the clinical laboratory at each site. As many of these laboratory tests are commonly obtained for clinical purposes, these tests do not need to be repeated if a result is available from the clinical care of the participant within 2 hours of the time point (or within 12 hours of the T4 time-point).

In addition to traditional clinical markers, 25ml of blood will be obtained for future biomarker analysis (including inflammatory biomarkers, markers of endothelial function, and markers of mitochondrial function), and measurement of vitamin C, vitamin B1, and cortisol levels. Levels of vitamin C, vitamin B1, and cortisol will be measured at time T1 and time T3 only. 20ml of urine will be collected for future biomarker analysis at T1, T2, and T3.

If performed as part of standard-of-care, results of urinalysis and urine sediment testing will be collected prior to enrollment.

### 4.5.3 Biomarker tube initial processing and shipping

Please see accompanying blood collection standard operating procedure for full details. In brief, 15ml of blood will be drawn into EDTA tubes and 10ml of blood will be drawn into a corvac tube. From one of the EDTA tubes, 3ml of whole blood will be initially drawn and separated into 3x 1ml aliquots. Plasma will then be isolated from the EDTA tube(s) and aliquoted into cryovials as follows: 2x 1ml aliquots and the remainder in 0.5ml aliquots. Serum will then be isolated from the corvac tube, and separated into 1ml aliquots. Cryovials will be protected from light and frozen at -80°C until processing. An additional 20ml of urine will also be collected, centrifuged, and separated into 1ml aliquots then frozen at -80°C until processing.

 Sites will be expected to ship frozen samples to the coordinating center after every 5 enrollments. The coordinating center will assist with all shipping procedures.

### 4.6 Study flow diagram



### 4.7 General Sepsis Management

Investigators should follow local sepsis management guidelines. No specific sepsis bundle is required by this study, however the early administration of antibiotics, maintenance of a mean arterial pressure ≥65mmHg with a combination of volume resuscitation and vasopressors, and early source control are recommended—as detailed in the Suriving Sepsis Guidelines.<sup>55</sup> Elements of sepsis care should be reported on the online case report form (CRF).

### 4.8 Glucometer use during the study period

High dose vitamin C has been shown to falsely elevate glucose level readings when measured with certain point-of-care glucometers employing glucosedehydrogenase-pyrroloquinoline quinone amperometric methods<sup>56</sup>. Some commonly used glucometer brands using this approach include Accu-Chek (Roche Diagnostic) and Optium (Abbott Diabetes Care) (but not StatStrip; Nova Biomedical). While the effects of high-dose vitamin C on glucometer readings have been seen primarily at higher doses of vitamin C than are intended for use in this trial, <sup>56</sup> we recommend that sites explore what glocumeters are in use in local ICUs. If locally used glucometers may be impacted by high serum concentrations of vitamin C (as determined by the manufacturer), we recommend that clinical teams caring for enrolled participants be alerted to the possibility of falsely elevated blood-glucose levels when measured by glucometer. If there is a clinical concern about a glucose reading obtained via glucometer, a serum glucose should be obtained which will not be impacted by vitamin C. In the event of an emergency related to suspected hypoglycemia, glucose should be immediately given while a serum glucose level is pending.

#### 5. OUTCOMES

### 5.1 Definitions

### 5.1.1 Primary Outcome

The primary outcome will be the absolute change in the Sequential Organ Failure Assessment (SOFA]) score from enrollment (time=0) to 72 hours after drug administration. The SOFA score will be defined using a modification in which the SaO2/FiO2 ratio is substituted for the PaO2/FiO2 ratio

 as has been previously described.<sup>57</sup> This modified score will be used so that participants without an existing arterial catheter can be spared arterial puncture.

| Points | SaO2*/FiO2 <sup>§</sup> | Blood Pressure | GCS | Bilirubin<br>(mg/dL) | Creatinine<br>(mg/dL) | Platelets<br>(x10 <sup>3</sup> µL) |
|---|---|---|---|---|---|---|
| 1 | <512 | < 70 mm/Hg | 13–14 | 1.2–1.9 | 1.2 – 1.9 | <150 |
| 2 | <357 | dopamine ≤ 5 μg/kg/min or<br>dobutamine<br>(any dose) | 10–12 | 2–5.9 | 2.0 – 3.4 | <100 |
| 3 | <214 | dopamine > 5μg/kg/min,<br>epinephrine/norepinephrine<br>≤ 0.1 μg/kg/min | 6–9 | 6–11.9 | 3.5 - 4.9<br>Or<br>UOP <sup>†</sup> <500ml/day | <50 |
| 4 | <89 | dopamine > 15,<br>epinephrine/norepinephrine<br>> 0.1 μg/kg/min | <6 | >12 | > 5.0<br>UOP <sup>†</sup> <200ml/day | <20 |

\*SaO2=Oxygen saturation (%); § = Fraction of inspired oxygen (%); II = Glasgow Coma Scale; † = Urine Output

### 

### 5.1.2 Key Secondary Outcomes

<u>Incidence of Acute Renal Failure</u> – Renal failure will be defined as the development of Kidney Disease Improving Global Outcomes [KDIGO] Stage 3 acute kidney injury during the index ICU stay after study enrollment.<sup>58</sup>

| KDIGO Stage | Serum creatinine criteria | Urine output criteria |
|---|---|---|
| 1 | Increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.4 µmol/l) or increase to more than or equal to 150% to 200% (1.5-to 2-fold) from baseline | Less than 0.5 ml/kg per hour for more than 6 hours |
| 2 | Increase in serum creatinine to more than 200% to 300% (> 2- to 3- fold) from baseline | Less than 0.5 ml/kg per hour for more than 12 hours |
| 3 | Increase in serum creatinine to more than 300% (> 3-fold) from baseline (or serum creatinine of more than or equal to 4.0 mg/dl [≥ 354 µmol/l] with an acute increase of at least 0.5 mg/dl [44 µmol/l]) | Less than 0.3 ml/kg per hour for<br>24 hours or anuria for 12 hours<br>OR<br>New renal replacement therapy<br>(RRT) |

<u>30-Day Mortality</u> – Mortality at 30-days. This will be assessed by review of the medical records if the participant remains in the hospital or if the participant expired while in the hospital. If the participant was discharged, 30-day mortality will be assessed by contacting the participant by phone or by searching the National Center for Health Statistics (NCHS) National Death Index (NDI) consistent with a recent multicenter phase III trial in sepsis.<sup>23</sup> Phone calls will be made by the research team at each site.

#### **5.2 Rationale for Outcomes**

**Change in SOFA score:** Organ failure is highly associated with mortality<sup>59</sup> and improvement in organ function is a key goal for critical care physicians. In the study by Marik et al.<sup>36</sup>, participants who received the 3-drug regimen had substantial improvements in the trajectory of organ failure over the first 72-hours of their ICU stay. If the combination of vitamin C, hydrocortisone, and vitamin B1 can improve organ function in the first 72-hours following ICU admission, we believe that clinicians will likely quickly adopt this safe and inexpensive therapy. Importantly, this outcome can be measured early in the hospital stay and is therefore less likely to be affected by other potential elements of hospital care that can affect more distal outcomes (e.g., mortality).

**Kidney Injury:** Renal failure has been estimated to occur in 23% of participants with sepsis and over 50% of participants with septic shock. In studies of participants with septic shock, there is a step-wise increase in mortality with worsening acute kidney injury (AKI). In addition, many participants who experience renal injury during septic shock do not recover renal function prior to hospital discharge and may require long term dialysis. As both data from the study by Marik et. al. and a separate study of vitamin B1 in septic shock have shown substantial improvements in renal outcomes, kidney failure is a natural secondary outcome and one that could change practice independently from other factors – in other words, many clinicians would likely provide this therapy if they knew that kidney function could be protected, since this organ is vital to long-term health.

**Mortality:** Finally, we will measure 30-day mortality. We anticipate that the combination of vitamin C, hydrocortisone, and vitamin B1 will reduce mortality in this high-risk population.

### **5.3 Additional Secondary Outcomes**

1727 5.3.1 Additional secondary outcomes

Additional secondary outcomes will include length of ICU stay, length of hospital stay, ventilator-free days over the first 7-days after enrollment, shock-free days over the first 7-days after enrollment, and the incidence of delirium on day #3 of the ICU stay (as assessed using the Confusion Assessment Method [CAM-ICU] system). Sites at which the CAM-ICU is performed daily as part of standard-of-care should assess whether delirium occurs on any day during the initial ICU stay. See Appendix #2.

### 5.3.2 90-day follow-up for Quality of Life assessment

Sites may choose to participate in a long-term outcomes substudy exploring the effects of ascorbic acid, hydrocortisone, and thiamine vs. placebo on quality of life following sepsis. If a site chooses to participate, a trained research assistant/investigator at the site (who is blinded to treatment arm) will contact all participants who were alive at 30-days, and perform the SF-36 at day 90 following enrollment. The SF-36 is a 36-Item Short-Form Health Survey (SF-36), a validated survey of general quality of life in adults, can be administered in person or over the telephone by research personnel. It measures eight different dimensions: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions, as well as one question asking about perceived changes in health. The telephone version of the 36-Item Short-Form Health Survey has been validated<sup>63,64</sup> and used in sepsis. 65-68

### 5.4 Safety

5.4.1 Definitions

The following definitions will be used<sup>69</sup>:

<u>Adverse event</u>: any untoward medical occurrence in a participant to whom a medicinal product is administered and which does not necessarily have a causal relationship with this treatment

<u>Serious adverse event</u>: any untoward medical occurrence that at any dose requires inparticipant hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, results in a congenital anomaly or birth defect, is life-threatening, or results in death

<u>Unexpected serious adverse event</u>: a serious adverse reaction, the nature, severity or outcome of which is not consistent with the reference safety information

### 

### 5.4.2 Specific adverse event data collection

 To assess specific amd potentially serious adverse events that may be related to the combination of the study medications, we will collect data on the following:

| Serious Adverse Event | Definition |
|---|---|
| Hyperglycemia | Serum glucose >300mg/dl in the first 120-hours after |
| | enrollment |
| Hypernatremia | Serum sodium (> 150 mmol/L) occurring in the first 120- |
| | hours after enrollment |
| New Infection | As data made and levelle a site and a site of investigation of a set |
| Catheter-site | As determined by the site principal investigator at each site. Should be a new organism or site of infection and |
| Lung | believed to be unrelated to the initial presenting |
| Gastrointestinal | infectious source. Many will have the initiation of new |
| Urinary tract | antibiotics or a change in antibiotics. |
| Other | antibiotics of a change in antibiotics. |
| Serious allergic reaction | Anaphylaxis or other allergic reaction requiring systemic |
| - | corticosteroids. Allergic reaction should be related (or |
| | suspected to be related) to the study medicaiton |
| Renal calculus | Development of a renal calculus between enrollment |
| | and 30-day follow-up (based on question asked during |
| | follow-up phone call). |

### 

### 5.4.3 Adverse Event Reporting

the site investigator) will be reported to the and all above listed Serious Adverse Events will be reported to the coordinating site, the data safety monitoring board (see below), and the regulatory authorities as applicable (i.e. IRB, FDA). Reporting of Serious Adverse Events will be done in aggregate after every 50 patients are enrolled. Unexpected Serious Adverse Event will additionally

Any Unexpected Serious Adverse Events thought to be related to the study drug (as determined by

1773 be report

be reported to the coordinating site within 72-hours.

### 5.4.5 Safety Monitoring Labs

 As detailed above, safety monitoring labs will be obtained at 120-hours, after completion of the study protocol.

### 

### 6. SAMPLE SIZE CALCULATION AND STATISTICAL ANALYSIS PLAN

## **6.1 Sample size calculation** 1781 The study has been powered

The study has been powered to have at least 80% power for the primary outcome and all key secondary outcomes as follows:

**SOFA Score**: Based on preliminary data<sup>36</sup>, we conservatively anticipate a decrease in SOFA score of 6 (standard deviation [SD]: 4) in the treatment group and 4 (SD: 2) in the placebo group. With these estimates, enrollment of **200 participants (100/arm)** at an alpha of 0.05 and using a t-test with unequal variance, the trial will provide > 99% power to detect a statistical significant difference between groups.

 **Kidney Injury:** Based on preliminary data from our study of vitamin B1 in septic shock,<sup>38</sup> we anticipate that 30% of participants in the treatment group and 55% in the placebo group will have renal failure which will result in a 94% power for this outcome. This calculation and following calculation were performed using the Fisher's exact test.

**Mortality:** Based on preliminary data<sup>37,70,71</sup>, we anticipate that the control group will have a mortality of 40%. We estimate a treatment effect of 50% (risk ratio: 0.50) resulting in a mortality of 20% in the treatment group. With these estimates, 182 participants will lead to 80% power. To further increase the trial's power and due to potential loss-to-follow-up, we will aim to enroll 200 participants. These

estimates are conservative compared to the Marik et al. study which found a treatment effect corresponding to a risk ratio of 0.21 which persisted in adjusted analysis.<sup>36</sup>

# 6.2 Statistical analysis plan

6.2.1 General considerations

The statistical analyses and reporting will adhere to the CONSORT guidelines.<sup>72,73</sup> All tests will be two-sided, a p-value < 0.05 will be considered significant, and all confidence intervals will have 95% coverage. All analyses will be conducted on a modified intention-to-treat basis only including participants receiving at least the first dose of the study medications. In a double-blind trial, this approach is unbiased while increasing precision.<sup>74</sup> The two groups will be compared in relation to baseline characteristics using descriptive statistics.

The persons conducting the statistical analysis will be blinded to the randomized allocation. Groups will be designated as "A" and "B" until all pre-specified analyses are performed and shared with all authors and the Data Safety Monitoring Board.

#### 6.2.2 SOFA score and renal failure

The change in SOFA score will be calculated and compared between groups using the Wilcoxon Rank Sum test (if the change is not normally distributed) or by a t-test if the change is approximately normally distributed. Fisher's exact tests will be used to compare the incidence of renal failure during the index ICU stay.

 If a participant expires prior to the 72-hour time point, SOFA scores will be imputed based on a predefined plan as follows. If a participant expires before 24-hours has elapsed, a 20% increase from baseline will be imputed. If a participant expires between 24-hours and 48-hours, a 15% increase from the 24-hour time point will be imputed. If a participant dies between 48-hours and 72-hours, a 20% increase from the 24-hour time point will be imputed. Sensitivity analyses will be performed using various other imputation techniques. Specifically, we will perform 1) a sensitivity analysis in which the worst possible SOFA score (score of 24) is imputed for those participants who expire, 2) a sentivity analysis in which the last SOFA score for participants who expire will be carried forward, and 3) a sensitivity analyses were chosen to model 'worst-possible' and 'best-possible' scenarios. For the secondary outcome of renal failure, participants who expire during their ICU stay will be assessed to have developed renal failure if they demonstrated any degree of unresolved KDIGO acute kidney injury prior to death. If there was no evidence of acute kidney injury prior to death or if kidney injury had fully resolved, these participants will be assessed as not having developed renal failure.

#### 6.2.3 30-day mortality

Survival until 30 days will be analyzed using survival analysis. Participants lost to follow-up will be censored and the censoring will be assumed non-informative. Results will be presented with Kaplan-Meier curves and the groups compared using the log-rank test. Hazard ratios with 95% confidence intervals will be obtained using Cox's proportional hazards models. The proportional hazards assumption will be verified by visual inspection of the Kaplan-Meier curves and statistically by including a product term (i.e. "interaction") between the treatment group variable and the natural logarithm of time in the model. If the proportional hazards assumption is not met, only the Kaplan-Meier curves and the p-value from the log-rank test will be presented.

Adverse events and other binary outcomes will be presented and analyzed like renal failure.

### 6.2.4 Additional Secondary Analyses

Both ICU and hospital length of stay will be compared using Wilcoxon Rank Sum tests. Ventilator and shock free days over the first 7-days after enrollment will likewise be compared using the

Wilcoxon Rank Sum given that the data will likely be not normally distributed. In these latter two analyses, patients who expire prior to 7-days will be assessed to have 0 ventilator or shock free days if they had died while on a ventilator or vasopressor respectively. The incidence of delirium will be compared using the Fisher's exact test. For the quality-of-life outcome (i.e. 90-day SF-36), the primary analysis will only include patients with available data. As a secondary analysis, multiple imputation will be used to estimate SF-36 scores in all patients not known to be dead at 90 -days.

### 6.2.5 Subgroup analyses

The analysis will include three pre-defined subgroup analyses for the primary and key secondary outcomes according to 1) participants with initially high SOFA scores ( $\geq$ 9). This cut-off was chosen to represent a population with a  $\geq$ 50% predicted likelihood of mortality<sup>78</sup> 2) baseline vitamin B1 deficiency and 3) baseline adrenal insufficiency. We will not plan to perform a subgroup analysis according to vitamin C deficiency, as prior work has shown that the vast majority of participants with septic shock have vitamin C levels below the reference range. Witamin B1 deficiency will be defined as a plasma vitamin B1 level  $\leq$  7 nmol/L as has been previously described. Adrenal insufficiency will be defined as a cortisol level  $\leq$ 10 $\mu$ g/dL. The trial is not powered to detect subgroup differences and these will be considered exploratory and hypothesis generating.

### 6.2.6 Statistical stopping criteria

Since the primary outcome is not mortality, there will be no formal stopping criteria for efficacy. There will be no predefined stopping criteria for futility since enrollment of the full cohort might allow for detection of efficacy in subgroups or in other outcomes even if the primary outcome is negative.

#### 7. DATA COLLECTION AND MANAGEMENT

### 7.1 Data collection process

Data collection will be the responsibility of the individual site investigators with oversite from the trial coordinating center. Most variables (i.e. demographics, sepsis characteristics and laboratory results) will be obtained prospectively from the electronic medical record. 30-day follow-up regarding safety and mortality end-points will be obtained via telephone call post-discharge (unless the participant remains in the hospital at 30-days). Data will be entered directly into the online database software (see below).

#### 7.2 Variables

Will be provided on the online CRF. A PDF version is available upon request.

### 7.3 Data quality and validity

Data quality and validity will be optimized by using a detailed data dictionary which will be distributed to all sites. Data quality will be monitored both centrally by the coordinating site and locally by each site principal investigator.

#### 7.4 Data storage and security

The database application we will use is REDCap Cloud (https://www.redcapcloud.com/). REDCap Cloud is a professional database that provides a user-friendly interface. The REDCap Cloud data management system is secure, fully compliant with all regulatory guidelines, and includes a complete audit-trail for data entry validation. Through these mechanisms, as well as relevant training for all involved parties, participant confidentiality will be safeguarded. All members of the research team will be required to complete standardized training in REDCap cloud, which will be documented within the software.

The consent form and other trial documents for each participant will initially be stored in a secure, locked place at the individual sites. Participating sites will be responsible for maintaining their own trial documents and study materials (e.g. signed ICFs, site logs etc). Trial documents generated at the Coordinating Center will be maintained the Coordinating Center. Following completion of the

trial, documents will be maintained for a period of at least 2-years at each site per FDA regulations (or longer depending on local IRB guidelines).

### 8. ETHICAL CONSIDERATIONS

#### 8.1 Risks and Benefits

8.1.1 Potential benefits

**Potential Benefits to Individual Participant:** Assuming our hypothesis is correct and our results are comparable to those previously published<sup>36</sup>, individual participants enrolled in our study and randomized to the treatment arm will benefit from a better trajectory of organ failure and improved mortality. As many participants who survive an initial episode of sepsis will have a future admission for sepsis, participants participating in this study but randomized to the placebo arm may see a future benefit from knowledge gained.

**Potential Benefits to Society:** Septic shock remains a highly morbid clinical condition for which there is no specific therapy. Our study, assuming our hypothesis is confirmed, will provide strong support for the widespread adoption of vitamin C, corticosteroids, and vitamin B1 for participants with septic shock. This, in turn, will significantly improve participant outcomes and reduce the global burden of death related to septic shock. Thus, even if participants are randomized to the placebo arm, their involvement with this study has tremendous potential benefits for society as whole. If vitamin C, corticosteroids, and vitamin B1 are found to be neutral or harmful (the latter being highly unlikely), society will benefit as the study will likely prevent the widespread dissemination of an ineffective medication combination.

#### 8.1.2 Potential harms

## **Study Drug**

Vitamin C – Ascorbic acid is a water-soluble essential vitamin that is safe even at high doses. Nevertheless, adverse effects related to high-dose ascorbic acid have been described. These adverse effects include diarrhea/abdominal bloating, increased oxalate excretion, iron overload in participants with hemochromatosis, and hemolysis in participants with G6PD deficiency. We exclude participants with known renal failure (CKD  $\geq$ 3b), known G6PD deficiency, or known hemochromatosis to limit these potential risks. We will additionally exclude participants with known allergy to ascorbic acid. Ascorbic acid has additionally been used in at least 3 clinical trials in critically-ill populations without major associated adverse effect.

Hydrocortisone – Hydrocortisone is a well-established medication for the treatment of refractory shock in sepsis. Some studies (e.g. CORTICUS) have found an increased incidence of secondary infection in participants with septic shock who receive steroids. This finding has not been replicated in other large trials of corticosteroids for sepsis. Additional hypothetical risks to the administration of hydrocortisone to participants with septic shock (e.g. increased gastro-intestinal bleeding, muscle weakness, and delirium) have not been found in clinical trials of corticosteroids in sepsis. In Interest Principal sepsis (e.g. increased gastro-intestinal bleeding, muscle weakness, and delirium) have not been found in clinical trials of corticosteroids in sepsis. In Interest Principal sepsis (e.g. increased gastro-intestinal bleeding, muscle weakness, and delirium) have not been found in clinical trials of corticosteroids in sepsis. In Interest Principal sepsis (e.g. increased gastro-intestinal bleeding, muscle weakness, and delirium) have not been found in clinical trials of corticosteroids in sepsis.

Hydrocortisone will not be tapered in this study as prior studies have shown benefit with corticosteroids in septic shock without a taper. <sup>80</sup> In addition, a recent large trial of corticosteroids in septic shock (ADRENAL, NEJM 2018) randomized patients to 7-days of corticosteroids or placebo and did not include a taper. In that trial there was no reported difference in rates of recurrent shock.

Vitamin B1 – The only potential serious side effect that has been reported from vitamin B1 administration is an extremely rare anaphylactic reaction (1:250,000 cases) and this might not even be of issue with the current manufactured version of vitamin B1 in the United States. The risk of an anaphylactic reaction was associated with a vitamin complex dispensed in Europe, and whether

vitamin B1 was the actual offending agent remains unknown; however, this 0.0004% theoretical chance of an adverse reaction is incredibly low. In a series of 989 participants in the United States who received intravenous vitamin B1, none had an anaphylactic reaction and the only reported side effects were minor consisting of transient local irritation or in one case pruritus (0.093%). Further safety data comes from the clinical use of intravenous vitamin B1 at our coordinating site. At Beth Israel Deaconess Medical Center (BIDMC, coordinating center) vitamin B1 is provided liberally for participants with nutritional deficiency – for example, BIDMC has administered intravenous vitamin B1 in over 8,000 separate participant encounters from 2002 until present. Despite this heavy usage, no adverse reactions were reported in any of the 8,000 participant encounters.

The combination of vitamin C, hydrocortisone and vitamin B1 – To date, the only study of the combination of vitamin C, hydrocortisone and vitamin B1 was the above referenced study by Marik et. al.

 All procedures will take place at the study site. All research procedures and monitoring will be conducted by experienced personnel, and participants will be in the ICU given critical illness. This permits closer observation and more detailed monitoring by clinicians familiar with the care of participants experiencing and resuscitated from septic shock.

#### **Blood Collection**

Most participants will have existing venous or arterial catheters in place and we will be able to collect blood from these ports, essentially eliminating the risks associated with blood collection. In the very rare case that a participant does not have an indwelling line, the risk of venipuncture is extremely low, and will not exceed the risk of clinical blood draws the participant will already be receiving.

### **Loss of Confidentiality**

All measures will be taken to ensure that no confidential information is released. All participant information will be stored in a password protected database to which only study investigators will have access. Additionally, all hard copies of study data will be kept in a locked office accessible only to study investigators. Thus, the risk of loss of confidentiality is very low.

### 9. MONITORING

### 9.1 Institutional Review Board (IRB)

The study will be reviewed and approved by the IRB at each participating site.

#### 9.2 Data Safety and Monitoring Board (DSMB)

The DSMB will be responsible for safeguarding the interests of trial participants, assessing the safety and efficacy of the interventions during the trial, and for monitoring the overall conduct of the clinical trial. The DSMB will consist of three clinicians with critical care experience in the management of septic participants. An independent biostatistician/epidemiologist will prepare all DSMB reports. The DSMB members will be chosen such to avoid any financial or intellectual conflicts of interest. The DSMB will review deidentified data after every 50 participants are enrolled to assess for safety; unless there are group differences necessitating unblinding (as determined by the DSMB), the DSMB will be blinded to treatment groups. The trial will continue while the DSMB review data. After each review, the DSMB will create a short report to the steering committee with recommendations for continuation, modifications, or termination of the trial. Criteria for recommending termination will be at the discretion of the DSMB and there will be no formal statistical criteria for termination due to efficacy or safety. A detailed charter for the DSMB will be provided.

#### **DSMB Members**

2007 Clifton Callaway, MD, PhD [DSMB Chair] University of Pittsburgh 2008 2009 400A Iroquois Pittsburgh, PA 15260 2010 (412) 647-8287 2011 callawaycw@upmc.edu 2012 2013 Professor (tenured) of Emergency Medicine; Executive Vice-Chair of Emergency Medicine; UPMC Professor of Emergency Medicine Research 2014 2015 **Expertise: Cardiac Arrest/Clinical Trials** 2016 2017 Taylor Thompson, MD Massachusetts General Hospital 2018 55 Fruit Street 2019 2020 Boston, MA 02114 (617) 724-7823 2021 tthompson1@partners.org 2022 Professor of Medicine, Harvard Medical School 2023 Director, Critical Care Translational Research, Pulmonary/Critical Care Unit, MGH 2024 2025 Medical Director, ARDS Network Clinical Coordinating Center 2026 Expertise: Sepsis/Clinical Trials 2027 2028 Shahzad Shaefi, MD MPH 2029 Beth Israel Deaconess Medical Center 2030 One Deaconess Raod 2031 Boston, MA 02115 2032 (617) 355-6286 sshaefi@bidmc.harvard.edu 2033 2034 Attending Physician, Department of Anesthesia, Critical Care and Pain 2035 Expertise: Critical Care Medicine 2036 2037 Manya Harsch, MS Principal Statistician, Technomics Research, LLC 2038 2039 (763) 473-6374 mharsch@technomicsresearch.com 2040 **Expertise: Biostatistics** 2041 2042 2043 **10 CLINICAL MONITORING PLAN** 

The detailed clinical monitoring plan has been developed and is available from the Coordianting

2044

2045

Center upon request.

#### 11. TIMELINE AND ENROLLMENT

### 11.1 Timeline



### 11.2 Screening & Enrollment

Enrollment at each site will be continuously monitored by the site investigator and the principal investigator. Each site will be expected to maintain a screening log including all participants who meet all eligibility criteria at that site. A standardized screening log will be provided to each site via RedCap Cloud—thus allowing for continuous updating of the screening log and will allow capture of all screening failures.

Enrollment will be competitive (i.e. without specific enrollment caps). Number of enrollments at each site will be shared with all sites on a monthly basis. Sites will be expected to complete all elements of the online CRF within 48-hours of each time point. In the case that a site continuously underperforms despite troubleshooting and feedback, the steering committee will evaluate whether enrollment will continue at that site.

#### 12. FUNDING

Funding for the present trial is provided by the Good Ventures Foundation (http://www.goodventures.org/). The funding agency will have no role in the design and conduct of the study, collection, management, analysis, and interpretation of the data, preparation, review, or approval of the manuscript, or the decision to submit the manuscript for publication.

#### 13. PUBLICATION

The manuscript will adhere to the CONSORT guidelines.<sup>72,73</sup> The principal investigator will be responsible for assigning authorship position and will follow authorship guidelines from the International Committee of Medical Journal Editors.<sup>82</sup> At a minimum, all members of the Steering Committee and all site Principal Investigators (for sites enrolling at least 10 participants) will be included in the primary author list. The main results will be presented at an international conference. The trial results will be shared with participating sites and via press releases but not directly with the participants.

#### 14. DATA SHARING

Six months after the publication of the last results, all de-identified individual participant data will be made available for data sharing. Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data. There will be no predetermined end date for the data sharing. Data will be available for any research purpose to all interested parties who have approval from an independent ethics review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Interested parties will be able to request the data by contacting the principal investigator. Authorship of publications emerging from the shared data will follow standard authorship guidelines from the International Committee of Medical Journal Editors<sup>82</sup> and might or might not include authors from the steering committee depending on the nature of their involvement.

#### 15. TASKS AND RESPONSIBILITIES

<u>Principal investigator and sponsor</u>: Overall responsibility for protocol development, funding, budget overview, data dictionary development, ethical approval, trial registration, daily management, trial oversight and collection of adverse events, contact to the pharmacy, contact to Good Clinical Practice monitoring unit and the data and safety monitoring board, assessment of overall recruitments, potential recruitment of additional sites, data analysis, and dissemination and presentation of results.

<u>Steering committee</u>: Protocol development, funding, budget overview, data dictionary development, trial oversight, dissemination of results, responsibilities as principal investigator for short time periods.

<u>Site investigators</u>: Responsible for site-specific enrollment, evaluation of eligible patients not included, education of personnel at participating sites, reporting of site-specific issues or challenges to the principal investigator, participant consent for data collection, collecting and reporting data regarding adverse drug events.

Clinical team: Administration of the study drug, participant consent for data collection.

#### 2108 References

- 2109 1. ICH Harmonised Tripartite Guideline. Integrated Addendum To ICH E6(R1): Guideline For Good Clinical Practice E6(R2). 2016;
- http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E6/E6\_R2\_\_Step \_\_4.pdf. Accessed June 30, 2017.
- 2. ICH Harmonised Tripartite Guideline. General Considerations for Clinical Trials E8. 1997;
- http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E8/Step4/E8\_Guideline.pdf. Accessed June 30, 2017.
- 2116 3. ICH Harnomised Tripartite Guidelines. Statistical Principles for Clinical Trials. 1998;
- http://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E9/Step4/E9\_Guideline.pdf. Accessed June 30, 2017.
- 2119 4. Chan AW, Tetzlaff JM, Altman DG, et al. SPIRIT 2013 statement: defining standard protocol items for clinical trials. *Ann Intern Med.* 2013;158(3):200-207.
- 5. Chan AW, Tetzlaff JM, Gotzsche PC, et al. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. *BMJ*. 2013;346:e7586.
- Fleischmann C, Scherag A, Adhikari N, et al. Global burden of sepsis: a systematic review (abstract).

  Critical Care. 2015;19 (suppl 1).
- 2125 7. Liu V, Escobar GJ, Greene JD, et al. Hospital deaths in patients with sepsis from 2 independent cohorts. *Jama*. 2014;312(1):90-92.
- 2127 8. Cohen J, Vincent JL, Adhikari NK, et al. Sepsis: a roadmap for future research. *The Lancet Infectious diseases*. 2015;15(5):581-614.
- 2129 9. Dellinger RP, Levy MM, Rhodes A, et al. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. *Critical care medicine*. 2013;41(2):580-637.
- Yende S, Linde-Zwirble W, Mayr F, Weissfeld LA, Reis S, Angus DC. Risk of cardiovascular events in survivors of severe sepsis. *American journal of respiratory and critical care medicine*.
   2133 2014;189(9):1065-1074.
- 2134 11. Mayr FB, Yende S, Angus DC. Epidemiology of severe sepsis. Virulence. 2014;5(1):4-11.
- 2135 12. Wintermann GB, Brunkhorst FM, Petrowski K, et al. Stress Disorders Following Prolonged Critical
   2136 Illness in Survivors of Severe Sepsis. *Critical care medicine*. 2015.
- 2137 13. Goodwin AJ, Rice DA, Simpson KN, Ford DW. Frequency, cost, and risk factors of readmissions among severe sepsis survivors. *Critical care medicine*. 2015;43(4):738-746.
- 2139 14. Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. *Jama*. 2010;304(16):1787-1794.
- 2141 15. Ortego A, Gaieski DF, Fuchs BD, et al. Hospital-based acute care use in survivors of septic shock. 2142 *Critical care medicine*. 2015;43(4):729-737.
- 2143 16. Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. *The New England journal of medicine*. 2003;348(16):1546-1554.
- 2145 17. Gaieski DF, Edwards JM, Kallan MJ, Carr BG. Benchmarking the incidence and mortality of severe sepsis in the United States. *Critical care medicine*. 2013;41(5):1167-1174.
- 2147 18. Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. *Critical care medicine*. 2001;29(7):1303-1310.
- 2150 19. Deans KJ, Haley M, Natanson C, Eichacker PQ, Minneci PC. Novel therapies for sepsis: a review. *The Journal of trauma*. 2005;58(4):867-874.
- 20. Eichacker PQ, Parent C, Kalil A, et al. Risk and the efficacy of antiinflammatory agents: retrospective and confirmatory studies of sepsis. *American journal of respiratory and critical care medicine*. 2002;166(9):1197-1205.
- 21. Opal SM, Dellinger RP, Vincent JL, Masur H, Angus DC. The next generation of sepsis clinical trial designs: what is next after the demise of recombinant human activated protein C?\*. *Critical care medicine*. 2014;42(7):1714-1721.

- 2158 22. Angus DC. The search for effective therapy for sepsis: back to the drawing board? *Jama*. 2011;306(23):2614-2615.
- 23. ProCess Investigators, Yealy DM, Kellum JA, et al. A randomized trial of protocol-based care for early septic shock. *The New England journal of medicine*. 2014;370(18):1683-1693.
- 24. Investigators A, Group ACT, Peake SL, et al. Goal-directed resuscitation for patients with early septic shock. *The New England journal of medicine*. 2014;371(16):1496-1506.
- 25. Mouncey PR, Osborn TM, Power GS, et al. Trial of early, goal-directed resuscitation for septic shock.

  The New England journal of medicine. 2015;372(14):1301-1311.
- 26. Asfar P, Meziani F, Hamel JF, et al. High versus low blood-pressure target in patients with septic shock. *The New England journal of medicine*. 2014;370(17):1583-1593.
- 27. Caironi P, Tognoni G, Masson S, et al. Albumin replacement in patients with severe sepsis or septic shock. *The New England journal of medicine*. 2014;370(15):1412-1421.
- 28. Holst LB, Haase N, Wetterslev J, et al. Lower versus higher hemoglobin threshold for transfusion in septic shock. *The New England journal of medicine*. 2014;371(15):1381-1391.
- 29. Abraham E, Anzueto A, Gutierrez G, et al. Double-blind randomised controlled trial of monoclonal antibody to human tumour necrosis factor in treatment of septic shock. NORASEPT II Study Group. *Lancet*. 1998;351(9107):929-933.
- 2175 30. Abraham E, Naum C, Bandi V, et al. Efficacy and safety of LY315920Na/S-5920, a selective inhibitor of 14-kDa group IIA secretory phospholipase A2, in patients with suspected sepsis and organ failure.

  2177 Critical care medicine. 2003;31(3):718-728.
- 2178 31. Abraham E, Wunderink R, Silverman H, et al. Efficacy and safety of monoclonal antibody to human tumor necrosis factor alpha in patients with sepsis syndrome. A randomized, controlled, double-blind, multicenter clinical trial. TNF-alpha MAb Sepsis Study Group. *JAMA : the journal of the American Medical Association*. 1995;273(12):934-941.
- 2182 32. Fisher CJ, Jr., Agosti JM, Opal SM, et al. Treatment of septic shock with the tumor necrosis factor receptor:Fc fusion protein. The Soluble TNF Receptor Sepsis Study Group. *The New England journal of medicine*. 1996;334(26):1697-1702.
- 2185 33. Bernard GR, Wheeler AP, Russell JA, et al. The effects of ibuprofen on the physiology and survival of patients with sepsis. The Ibuprofen in Sepsis Study Group. *The New England journal of medicine*. 1997;336(13):912-918.
- 2188 34. Marti-Carvajal AJ, Sola I, Gluud C, Lathyris D, Cardona AF. Human recombinant protein C for severe sepsis and septic shock in adult and paediatric patients. *The Cochrane database of systematic* reviews. 2012;12:CD004388.
- 2191 35. Ranieri VM, Thompson BT, Barie PS, et al. Drotrecogin alfa (activated) in adults with septic shock.
  2192 The New England journal of medicine. 2012;366(22):2055-2064.
- Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C and Thiamine
   for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. *Chest.* 2016.
- 2196 37. Donnino MW, Andersen LW, Chase M, et al. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. *Crit Care Med.* 2016;44(2):360-2198 367.
- 2199 38. Moskowitz A, Andersen LW, Cocchi MN, Karlsson M, Patel PV, Donnino MW. Thiamine as a Renal 2200 Protective Agent in Septic Shock. A Secondary Analysis of a Randomized, Double-Blind, Placebo-2201 controlled Trial. *Annals of the American Thoracic Society*. 2017;14(5):737-741.
- Teng J, Pourmand A, Mazer-Amirshahi M. Vitamin C: The next step in sepsis management? *J Crit Care*. 2017;43:230-234.
- Fowler AA, 3rd, Syed AA, Knowlson S, et al. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. *Journal of translational medicine*. 2014;12:32.

- Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. *Archives of surgery (Chicago, III : 1960)*. 2000;135(3):326-331.
- Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's
   requirement in septic shock. *Journal of research in pharmacy practice*. 2016;5(2):94-100.
- 43. Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y. Corticosteroids for treating sepsis.
   2212 Cochrane Database Syst Rev. 2015(12):CD002243.
- 2213 44. May JM, Harrison FE. Role of vitamin C in the function of the vascular endothelium. *Antioxidants & redox signaling*. 2013;19(17):2068-2083.
- Han M, Pendem S, Teh SL, Sukumaran DK, Wu F, Wilson JX. Ascorbate protects endothelial barrier function during septic insult: Role of protein phosphatase type 2A. *Free radical biology & medicine*. 2010;48(1):128-135.
- 2218 46. Sprung CL, Annane D, Keh D, et al. Hydrocortisone therapy for patients with septic shock. *The New England journal of medicine*. 2008;358(2):111-124.
- 47. Keh D, Trips E, Marx G, et al. Effect of Hydrocortisone on Development of Shock Among Patients
   With Severe Sepsis: The HYPRESS Randomized Clinical Trial. *Jama*. 2016;316(17):1775-1785.
- 2222 48. Okamoto K, Tanaka H, Makino Y, Makino I. Restoration of the glucocorticoid receptor function by the 2223 phosphodiester compound of vitamins C and E, EPC-K1 (L-ascorbic acid 2-[3,4-dihydro-2,5,7,8-2224 tetramethyl-2-(4,8,12-trimethyltridecyl)-2H-1-benzopyran-6 -yl hydrogen phosphate] potassium 2225 salt), via a redox-dependent mechanism. *Biochemical pharmacology*. 1998;56(1):79-86.
- 49. Fujita I, Hirano J, Itoh N, Nakanishi T, Tanaka K. Dexamethasone induces sodium-dependant vitamin
   C transporter in a mouse osteoblastic cell line MC3T3-E1. *The British journal of nutrition*.
   2001;86(2):145-149.
- Donnino MW, Andersen LW, Chase M, et al. Randomized, Double-Blind, Placebo-Controlled Trial of
   Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. *Critical care medicine*.
   2016;44(2):360-367.
- Gioda CR, de Oliveira Barreto T, Primola-Gomes TN, et al. Cardiac oxidative stress is involved in heart
   failure induced by thiamine deprivation in rats. *American journal of physiology Heart and circulatory* physiology. 2010;298(6):H2039-2045.
- Pacal L, Tomandl J, Svojanovsky J, et al. Role of thiamine status and genetic variability in
   transketolase and other pentose phosphate cycle enzymes in the progression of diabetic
   nephropathy. Nephrology, dialysis, transplantation: official publication of the European Dialysis and
   Transplant Association European Renal Association. 2011;26(4):1229-1236.
- 53. Kernan WN, Viscoli CM, Makuch RW, Brass LM, Horwitz RI. Stratified randomization for clinical trials.
   J Clin Epidemiol. 1999;52(1):19-26.
- Johnson K, Posner SF, Biermann J, et al. Recommendations to improve preconception health and health care--United States. A report of the CDC/ATSDR Preconception Care Work Group and the Select Panel on Preconception Care. MMWR Recommendations and reports: Morbidity and mortality weekly report Recommendations and reports. 2006;55(Rr-6):1-23.
- 2245 55. Rhodes A, Evans LE, Alhazzani W, et al. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. *Critical care medicine*. 2017;45(3):486-552.
- Flannery AH, Bastin MLT, Magee CA, Bensadoun ES. Vitamin C in Sepsis: When It Seems Too Sweet, It Might (Literally) Be. *Chest.* 2017;152(2):450-451.
- 2249 57. Pandharipande PP, Shintani AK, Hagerman HE, et al. Derivation and validation of Spo2/Fio2 ratio to impute for Pao2/Fio2 ratio in the respiratory component of the Sequential Organ Failure Assessment score. *Critical care medicine*. 2009;37(4):1317-1321.
- Mehta RL, Kellum JA, Shah SV, et al. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. *Critical care (London, England)*. 2007;11(2):R31.

- de Grooth HJ, Geenen IL, Girbes AR, Vincent JL, Parienti JJ, Oudemans-van Straaten HM. SOFA and mortality endpoints in randomized controlled trials: a systematic review and meta-regression analysis. *Crit Care.* 2017;21(1):38.
- Schrier RW, Wang W. Acute renal failure and sepsis. *The New England journal of medicine.* 2004;351(2):159-169.
- 2259 61. Kellum JA, Chawla LS, Keener C, et al. The Effects of Alternative Resuscitation Strategies on Acute 2260 Kidney Injury in Patients with Septic Shock. *American journal of respiratory and critical care* 2261 *medicine*. 2016;193(3):281-287.
- Ely EW, Inouye SK, Bernard GR, et al. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). *Jama*. 2001;286(21):2703-2710.
- Watson EK, Firman DW, Baade PD, Ring I. Telephone administration of the SF-36 health survey:
   validation studies and population norms for adults in Queensland. *Aust N Z J Public Health*.
   1996;20(4):359-363.
- Garcia M, Rohlfs I, Vila J, et al. Comparison between telephone and self-administration of Short Form Health Survey Questionnaire (SF-36). *Gac Sanit*. 2005;19(6):433-439.
- Schmidt K, Worrack S, Von Korff M, et al. Effect of a Primary Care Management Intervention on
   Mental Health-Related Quality of Life Among Survivors of Sepsis: A Randomized Clinical Trial. *Jama*.
   2016;315(24):2703-2711.
- 2273 66. Dinglas VD, Hopkins RO, Wozniak AW, et al. One-year outcomes of rosuvastatin versus placebo in sepsis-associated acute respiratory distress syndrome: prospective follow-up of SAILS randomised trial. *Thorax.* 2016;71(5):401-410.
- Zhang K, Mao X, Fang Q, et al. Impaired long-term quality of life in survivors of severe sepsis:
   Chinese multicenter study over 6 years. *Anaesthesist*. 2013;62(12):995-1002.
- Wittbrodt P, Haase N, Butowska D, et al. Quality of life and pruritus in patients with severe sepsis resuscitated with hydroxyethyl starch long-term follow-up of a randomised trial. *Crit Care.* 2013;17(2):R58.
- The European Parliament and the Council of the European Unit. Clinical Trials Regulation (CTR) EU
  No 536/2014. 2014; https://ec.europa.eu/health/sites/health/files/files/eudralex/vol1/reg 2014 536/reg 2014 536 en.pdf. Accessed July 18, 2017.
- Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine
   for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. *Chest*.
   2017;151(6):1229-1238.
- Rhee C, Dantes R, Epstein L, et al. Incidence and Trends of Sepsis in US Hospitals Using Clinical vs Claims Data, 2009-2014. *JAMA*. 2017;318(13):1241-1249.
- Schulz KF, Altman DG, Moher D, Group C. CONSORT 2010 statement: updated guidelines for
   reporting parallel group randomised trials. *BMJ*. 2010;340:c332.
- 73. Moher D, Hopewell S, Schulz KF, et al. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. *BMJ.* 2010;340:c869.
- Fergusson D, Aaron SD, Guyatt G, Hebert P. Post-randomisation exclusions: the intention to treat principle and excluding patients from analysis. *BMJ.* 2002;325(7365):652-654.
- Fleming T, Harrington D. Nonparametric estimation of the survival distribution in censored data. *Communications in Statistics Theory and Methods.* 1984;13(20):2469–2486.
- 2297 76. Cox D. Regression models and life tables. *Journal of the Royal Statistical Society.* 1972;Series B(20):187–220.
- 2299 77. Kleinbaum D, Klein M. Survival Analysis: A Self-Learning Text. 3rd ed: Springer; 2013.
- 78. Vincent JL, de Mendonca A, Cantraine F, et al. Use of the SOFA score to assess the incidence of organ
   dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working
- group on "sepsis-related problems" of the European Society of Intensive Care Medicine. *Critical care medicine*. 1998;26(11):1793-1800.

| 2304 | 79. | Levine M, Rumsey SC, Daruwala R, Park JB, Wang Y. Criteria and recommendations for vitamin C |
|---|---|---|
| 2305 | | intake. <i>Jama</i> . 1999;281(15):1415-1423. |

- Annane D, Sebille V, Charpentier C, et al. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. *Jama*. 2002;288(7):862-871.
- Wrenn KD, Murphy F, Slovis CM. A toxicity study of parenteral thiamine hydrochloride. *Annals of emergency medicine*. 1989;18(8):867-870.
- 2310 82. International Committee of Medical Journal Editors. Defining the Role of Authors and Contributors.
  2311 2017; http://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role2312 of-authors-and-contributors.html. Accessed July 6, 2017.
- Taichman DB, Sahni P, Pinborg A, et al. Data Sharing Statements for Clinical Trials A Requirement of the International Committee of Medical Journal Editors. *N Engl J Med.* 2017;376(23):2277-2279.

| 2315 | Appendices |
|---|---|
| 2316 | Among div. A. Alabagasisticas |
| 2317 | Appendix 1: Abbreviations ICHInternational Conference on Harmonization |
| 2318<br>2319 | SPIRITStandard Protocol Items: Recommendations for Interventional Trials |
| 2319 | |
| 2320 | ACTAscorbic Acid, Corticosteroids, and Thiamine |
| | CKDChronic Kidney Disease SOFASequential Organ Failure Assessment |
| 2322 | INDInvestigational New Drug |
| 2323<br>2324 | FDAFood and Drug Administration |
| 2324 | ICUIntensive Care Unit |
| 2325 | |
| | SaO2Oxygen Saturation |
| 2327 | FiO2Fraction of Inspired Oxygen |
| 2328<br>2329 | GCSGlasgow Coma Scale |
| | UOPUrine Output RRTRenal Replacement Therapy |
| 2330<br>2331 | CAMConfusion Assessment Method |
| | NCHS National Center for Health Statistics |
| 2332<br>2333 | NDINational Death Index |
| 2333 | |
| 2334 | AKIAcute Kidney Injury SDtandard deviation |
| 2335 | |
| | CRFCase Report Form |
| 2337 | BIDMCBeth Israel Deaconess Medical Center (Coordinating Center) IRBInstitutional Review Board |
| 2338 | |
| 2339 | DSMBData Safety and Monitoring Board |
| 2340 | |
| 2341 | |
| 2342 | |
| 2343 | |
| 2344 | |
| 2345 | |
| 2346 | |
| 2347 | |
| 2348 | |
| 2349 | |
| 2350 | |
| 2351 | |
| 2352 | |
| 2353 | |
| 2354 | |
| 2355 | |
| 2356 | |
| 2357 | |
| 2358 | |
| 2359 | |
| 2360 | |
| 2361 | |
| 2362 | |

# **CAM-ICU Worksheet**

| Feature 1: Acute Onset or Fluctuating Course | Score | Check here if Present |
|---|---|---|
| Is the pt different than his/her baseline mental status? OR Has the patient had any fluctuation in mental status in the past 24 hours as evidenced by fluctuation on a sedation scale (i.e., RASS), GCS, or previous delirium assessment? | Either<br>question Yes<br>→ | |
| Feature 2: Inattention | | |
| <u>Letters Attention Test</u> (See training manual for alternate <b>Pictures</b> ) | | |
| <u>Directions</u> : Say to the patient, "I am going to read you a series of 10 letters. Whenever you hear the letter 'A,' indicate by squeezing my hand." Read letters from the following letter list in a normal tone 3 seconds apart. | Number of Errors >2 → | |
| SAVEAHAART | | |
| Errors are counted when patient fails to squeeze on the letter "A" and when the patient squeezes on any letter other than "A." | | |
| Feature 3: Altered Level of Consciousness | | |
| Present if the Actual RASS score is anything other than alert and calm (zero) | RASS<br>anything other<br>than zero → | |
| Feature 4:Disorganized Thinking | | |
| Yes/No Questions (See training manual for alternate set of questions) | | |
| <ol> <li>Will a stone float on water?</li> <li>Are there fish in the sea?</li> <li>Does one pound weigh more than two pounds?</li> <li>Can you use a hammer to pound a nail?</li> </ol> | Combined | |
| Errors are counted when the patient incorrectly answers a question. | number of | |
| <u>Command</u> Say to patient: "Hold up this many fingers" (Hold 2 fingers in front of patient) "Now do the same thing with the other hand" (Do not repeat number of fingers) *If pt is unable to move both arms, for 2 <sup>nd</sup> part of command ask patient to "Add one more finger" | errors >1→ | |
| An error is counted if patient is unable to complete the entire command. | | |

| Overall CAM-ICU | Criteria Met → | CAM-ICU Positive (Delirium Present) |
|---|---|---|
| Feature 1 plus 2 and either 3 or 4 present = CAM-ICU positive | Criteria Not Met → | CAM-ICU |
| | | Negative<br>(No Delirium) |

# 3. SUMMARY OF PROTOCOL CHANGES

| 2368<br>2369 | v2.1 – Original trial protocol. v1.0 of the protocol was a draft protocol that was updated following the |
|---|---|
| 2370 | initial investigator meeting. |
| 2371 | v2.2 – Added external study sites. Modifications to protocol at coordinating center (reflected in v2.3 |
| 2372 | for all sites). |
| 2373 | v2.3 – Change in exclusion criteria from CKD ≥3b [GFR < 45ml/hr]) to receiving renal replacement |
| 2374 | therapy. Clarification that sepsis should be the likely cause of hypotension resulting in vasopressor |
| 2375 | requirement and that consent/enrollment should be within 24-hours of meeting inclusion criteria. |
| 2376 | Change in contingency should open label thiamine be prescribed by the clinical tram. Allowance for |
| 2377 | a consideration of sample size adjustment should the SOFA score and/or mortality for the full study |
| 2378 | cohort (examined without consideration of study group) fall below that anticipated in the power |
| 2379 | analysis. Clarification of adverse event reporting procedures. |
| 2380 | v2.4 – Addition of study site. Correction of oversight in exclusion criteria with respect to clinical |
| 2381 | ascorbic acid supplementation. Clarification of SOFA scale to assign a renal SOFA score of 4 if a |
| 2382 | patient is started on renal replacement therapy. |